205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

| | Statistical Arialysis Flan Americinent i Final |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A Phase IIa, open-label, controlled, mono-center study to evaluate the efficacy, immunogenicity and safety of GSK Biologicals' candidate malaria vaccines RTS,S/AS01 <sub>E</sub> and RTS,S/AS01 <sub>B</sub> administered as various dose schedules according to a 0, 1, 7-month or a 0, 7-month schedule in healthy malaria-naïve subjects aged 18-55 years. 205081 (MALARIA-092) |
| eTrack study number and<br>Abbreviated Title | 205081 (MALARIA-092) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Amendment 1 Final: 05-DEC-2018 |
| Co-ordinating author: | PPD / PPD (Statistician) |
| Reviewed by: | PPD (Clinical Research and Development Lead) PPD (Lead Scientific writer) PPD (Scientific writer) PPD (Regulatory Affair) PPD (SERM physician) PPD (SERM Scientist) PPD (CLS Manager) PPD (Lead statistical analyst) PPD (Lead statistician) PPD (Public disclosure) |
| Approved by: | PPD (Clinical Research and Development Lead) PPD (Lead Scientific writer) PPD (Lead statistical analyst) PPD (Lead statistician) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14April 2017)

# 205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | T OF A | BBREVIATIONS | 9 |
| 1. | DOCL | JMENT HISTORY | 11 |
| 2. | STUD | Y DESIGN | 12 |
| _ | 0D.IE | OTIV (5.0 | 4.5 |
| 3. | 0BJE | CTIVES | |
| | 3.1. | Primary objective | |
| | 3.2. | Secondary objectives | |
| | 0.2. | 3.2.1. Efficacy | |
| | | 3.2.2. Immunogenicity | |
| | | 3.2.3. Safety | |
| | 3.3. | Tertiary objectives | |
| | | 3.3.1. Immunogenicity | |
| 4. | ENDP | OINTS | 16 |
| | 4.1. | Primary endpoint | 16 |
| | | 4.1.1. Efficacy | |
| | 4.2. | Secondary endpoints | |
| | | 4.2.1. Efficacy | |
| | | 4.2.2. Immunogenicity | |
| | 4.0 | 4.2.3. Safety | |
| | 4.3. | Tertiary endpoints | |
| 5. | ΛΝΛΙ | YSIS SETS | 20 |
| J. | 5.1. | Definition | |
| | 5.1. | 5.1.1. Enrolled Set | |
| | | 5.1.2. Intent-to-treat set (ITTS) | |
| | | 5.1.3. Solicited Safety Set | |
| | | 5.1.4. Per-Protocol Set for analysis of immunogenicity and | |
| | | efficacy (PPS for analysis of immunogenicity and efficacy) | 20 |
| | | 5.1.5. Adapted Per-Protocol Set for analysis of efficacy (Adapted | |
| | | PPS for analysis of efficacy) | |
| | 5.2. | Criteria for eliminating data from Analysis Sets | 21 |
| | | 5.2.1. Elimination from ITTS | 21 |
| | | 5.2.2. Elimination from the Solicited Safety Set | 21 |
| | | 5.2.3. Elimination from the PPS for analysis of immunogenicity | - 4 |
| | | and efficacy | 21 |
| | | 5.2.3.1. Excluded subjects | 21 |
| | | 5.2.4. Elimination from the Adapted PPS for analysis of efficacy | |
| | 5.3. | 5.2.4.1. Excluded subjects | 23 |
| | J.J. | Important protocol deviations not leading to elimination from per-<br>protocol analysis set | 23 |
| 6 | CT A T | ISTICAL ANALYSES | 24 |
| 6. | 6.1. | STICAL ANALYSES Demography | |
| | 0.1. | Domography | 4 |

| | | | 205081 (MALA<br>Statistical Analysis Plan Amendme | |
|---|---|---|---|---|
| | | 6.1.1. | Analysis of demographics/baseline characteristics planned in the protocol | |
| | 6.2. | Exposure | 9 | |
| | 0.2. | 6.2.1. | Analysis of exposure planned in the protocol | |
| | 6.3. | | analysis | |
| | | 6.3.1. | Analysis of efficacy planned in the protocol | |
| | | 6.3.2. | Additional considerations | |
| | | | 6.3.2.1. Case definition | |
| | | | 6.3.2.2. Risk periods | |
| | 6.4. | | genicity analysis | 26 |
| | | 6.4.1. | Analysis of immunogenicity planned in the protocol | 26 |
| | 0.5 | 6.4.2. | Additional considerations | |
| | 6.5. | • | of safety | |
| | | 6.5.1.<br>6.5.2. | Analysis of safety planned in the protocol | 21 |
| | | 0.5.2. | Additional considerations | 30 |
| 7. | ANAL | /SIS INTE | ERPRETATION | 30 |
| 0 | COND | LICT OF | ANALVOEC | 24 |
| 8. | 8.1. | | ANALYSESe of analyses | |
| | 8.2. | | al considerations for interim analyses | |
| | 0.2. | Otationica | a considerations for interim analyses | |
| 9. | CHAN | GES FRC | DM PLANNED ANALYSES | 31 |
| 10. | LIST C | F FINAL | REPORT TABLES, LISTINGS AND FIGURES | 31 |
| 11. | ANNE | X 1 STAN | IDARD DATA DERIVATION RULE AND STATISTICAL | |
| | METH | ODS | | 32 |
| | 11.1. | Statistica | al Method References | 32 |
| | 11.2. | | d data derivationd data derivation | |
| | | 11.2.1. | | |
| | | 11.2.2. | Dose number | |
| | | 11.2.3. | Demography | |
| | | 11.2.4. | Immunogenicity | |
| | | 11.2.5. | Safety | 34 |
| 12. | ANNE | X 2: TABL | LES, FIGURES AND LISTINGS | 37 |
| | 12.1. | Demogra | aphics & baseline characteristics | 37 |
| | 12.2. | Efficacy. | | 38 |
| | 12.3. | | genicity | |
| | 12.4. | | enicity and Safety | |
| | 12.5. | Individua | al data listings: | 46 |
| | 12.6. | | e of tables, figures AND LISTINGS | |
| | | 12.6.1. | Demographics and baseline characteristics | |
| | | 12.6.2. | Efficacy | |
| | | 12.6.3.<br>12.6.4. | ImmunogenicityReactogenicity and safety | |
| | | 14.0.7. | reading and salety | |

# 205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Intervals between study visits for the investigational vaccine groups: AduFx, 2PedFx, PedFx, and Adu2Fx | 13 |
| Table 2 | Intervals between study visits for the investigational vaccine group: Adu1Fx | 13 |
| Table 3 | Intervals between study visits for the infectivity control group | 13 |
| Table 4 | Toxicity grading scales for blood testing | 29 |

# 205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

# **LIST OF FIGURES**

| | | PAGE |
|----------|--------------|------|
| Figure 1 | Study design | 12 |

# 205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

# **LIST OF TEMPLATES**

| | | PAGE |
|---|---|---|
| Template 1 | Consort flow (Enrolled set) | 47 |
| Template 2 | Consort flow (Intent to treat set) | 47 |
| Template 3 | Summary of visit attendance (Intent-to treat set) | 48 |
| Template 4 | Summary of disposition <analysis name="" set=""></analysis> | 48 |
| Template 5 | Summary of important protocol deviations leading to elimination <analysis name="" set=""></analysis> | 49 |
| Template 6 | Deviations from protocol for age and intervals between study visits <analysis name="" set=""></analysis> | 50 |
| Template 7 | Summary of demographic characteristics <analysis name="" set=""></analysis> | 51 |
| Template 8 | Summary of demography and baseline characteristics <enrolled set=""></enrolled> | 52 |
| Template 9 | Summary of previous Hepatitis B vaccination (Intent-to-treat set) | 53 |
| Template 10 | Exposure to study vaccine by visit (Intent-to-treat) | 53 |
| Template 11 | Parasitemia incidence defined by a positive blood slide and vaccine efficacy versus control of <each group=""> (Per protocol set for analysis of immunogenicity and efficacy)</each> | 54 |
| Template 12 | Time to onset of parasitemia by blood slide (Per protocol set for analysis of immunogenicity and efficacy) | 55 |
| Template 13 | Cumulative incidence of parasitemia onset defined by positive blood slide for all groups (Per protocol set for analysis of immunogenicity and efficacy) | 55 |
| Template 14 | Number and percentage of subjects with <assay description=""> equal or above <cut-off> and GMCs (Per protocol set for analysis of immunogenicity and efficacy)</cut-off></assay> | 56 |
| Template 15 | Reverse cumulative distribution curve for <assay description=""> <timing> (Per protocol set for analysis of immunogenicity and efficacy)</timing></assay> | 57 |
| Template 16 | Comparison of the log-transformed means of the <anti-cs> antibodies <repeat c-term="" full-length=""> at post-vaccination of <each adufx="" non-protected="" protected="" schedule="" vaccination="" versus=""> (Per protocol set for analysis of immunogenicity and efficacy)</each></repeat></anti-cs> | 57 |
| | - , , | |

| | 20 | 5081 | (MALA | ٩RI | A-( | J92 |
|------|----|------|-------|-----|-----|-----|
| <br> | | - | | | | |

| Template 17 | Box and whiskers plot of <assay description=""> <timing> (Per protocol set for analysis of immunogenicity and efficacy)</timing></assay> | |
|---|---|---|
| Template 18 | Evolution over time for <assay (per="" analysis="" and="" descrition="" efficacy)<="" for="" immunogenicity="" of="" protocol="" set="" td=""><td>.58</td></assay> | .58 |
| Template 19 | Compliance in completing solicited adverse events information (intent-to-treat) | .59 |
| Template 20 | Incidence and nature of symptoms (solicited and unsolicited) within 7-day following each vaccination and overall (Intention-to-treat set) | .60 |
| Template 21 | Incidence of solicited <local general=""> symptoms within 7-day following each vaccination and overall (Intention-to-treat set)</local> | .61 |
| Template 22 | Incidence of temperature by maximum value, within 7 days following each vaccination and overall (Intention-to-treat set) | 62 |
| Template 23 | Summary of <subjects by="" followed="" vaccinations="" with=""> at least one <serious fatal="" related="" serious=""> unsolicited adverse events <medically attended="" visits="">, <within 30="" any="" days="" from="" of="" period="" post-challenge="" start="" study="" to="" vaccination="" within=""> (Intention-to-treat set)</within></medically></serious></subjects> | . 63 |
| Template 24 | Summary of occurrences and subjects with at least one serious unsolicited adverse events from study start until last study visit (D314) (Intention-to-treat set) | .63 |
| Template 25 | Summary of subjects by unsolicited event category, <within 30="" any="" days="" from="" of="" period="" post-challenge="" start="" study="" to="" vaccination="" within=""> (Intention-to-treat set)</within> | .64 |
| Template 26 | Listing of potential immune-mediated disorders (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment (Intent to treat set) | .64 |
| Template 27 | Listing of SAEs reported from study start to 28 days post challenge (Intention-to-treat set) | .64 |
| Template 28 | Listing of (S) AEs and solicited symptoms leading to study/treatment discontinuation (Intent to treat set) | .65 |
| Template 29 | Summary of hematology and biochemistry results (Intention-to-treat set) | .65 |
| Template 30 | Summary of subjects taking a concomitant medication with <7 days following each vaccination and overall / during challenge phase> (Intent to treat set) | .65 |

| Template 31 Bar graph of the daily prevalence of <pain redness="" swelling=""> between day 1 and day 7 following each vaccination (Intent to treat set) 66</pain> | |
|---|---|
| | between day 1 and day 7 following each vaccination (Intent to |
| Template 32 | |

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

### LIST OF ABBREVIATIONS

AE Adverse event

ALT Alanine aminotransferase

Anti-CS Antibody to the *Plasmodium falciparum* circumsporozoite (CS) repeat

domain

Anti-HBs Antibody to the hepatitis B surface antigen

AS01<sub>B</sub> GSK's proprietary Adjuvant System containing MPL, QS-21 and

liposome (50 µg MPL and 50 µg QS-21)

AS01<sub>E</sub> GSK's proprietary Adjuvant System containing MPL, QS-21 and

liposome (25 µg MPL and 25 µg QS-21)

AST Aspartate aminotransferase

ATP According-To-Protocol

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

CLS Clinical laboratory sciences

CRF Case Report Form

C-term CS terminal portion of the protein

CTRS Clinical Trial Registry Summary

eCRF electronic Case Report Form

EPT Endpoint titer

ES Exposed Set

EU/ml ELISA unit per milliliter

GMC Geometric mean concentration

GSK GlaxoSmithKline

HBsAg Hepatitis B surface Antigen

ICH Internal Conference on Harmonization

IgG Immunoglobulin G

IU/ml International units per milliliter

ITTS Intent-To-Treat Set

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

mIU/ml Milli International units per milliliter

NP Not protected

P Protected

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

PCR Polymerase chain reaction

PD Protocol Deviation

pIMD potential Immune Mediated Disease

PPS Per-Protocol Set

SAE Serious adverse event

SAS Statistical Analysis System

SAP Statistical Analysis Plan

SD Standard Deviation

SERM Safety Evaluation and Risk Management

SHS Study Headline Summary

TFL Tables Figures and Listings

TOC Table of Content

UL Upper Limit of the confidence interval

ULN Upper Limit of normal range

VE Vaccine Efficacy

WBC White blood cells

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 24-MAY-2018 | Final version | Administrative Change – 19-JUN-2017 |
| 05-DEC-2018 | Amendment 1: Addition of one analysis set and update in the standard computation rules | Administrative Change – 19-JUN-2017 |

# 2. STUDY DESIGN

Figure 1 Study design



D: Day; Mth: month; R: RTS,S; SCR: Screening; V: visit. \* Blood sample for estimation of subjects with parasitemia (PCR testing) will be collected on the day of subject entry into the hotel phase (Day 295 [Visit 16]); blood sample for biochemistry and hematology parameters will be collected the day of first parasitemia and blood sample for assessment of parasitemia (blood smear) will be collected daily for 14 days (from Day 291 [Visit 12] to Day 304 [Visit 25]) and then every two days for nine days (Day 306 [Visit 26], Day 308 [Visit 27], Day 310 [Visit 28], Day 312 [Visit 29], and Day 314 [Visit 30]).

05-DEC-2018 

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

The following table gives the intervals between study visits at defined visits to apply, as described in the protocol:

Table 1 Intervals between study visits for the investigational vaccine groups: AduFx, 2PedFx, PedFx, and Adu2Fx

| Interval | Optimal length of interval <sup>1</sup> | Allowed interval <sup>2</sup> |
|---|---|---|
| Visit 1 (Screening) → Visit 2 (1st vaccination) | 0 to 90 days | - |
| Visit 2 → Visit 3 (2 <sup>nd</sup> vaccination) | 28 days | $\pm$ 7 days |
| Visit 3 → Visit 5 | 7 days | ± 1 day |
| Visit 3 → Visit 6 | 30 days | $\pm$ 7 days |
| Visit 3 → Visit 7 (3 <sup>rd</sup> vaccination) | 168 days | ± 14 days |
| Visit 7 → Visit 9 | 7 days | ± 1 day |
| Visit 7 → Visit 10 | 30 days | $\pm$ 7 days |
| Visit 7 → Visit 11 (Challenge) | 90 days | + 14 days |
| Visit 11 → Visit 30 | 28 days | ± 7 days |
| Visit 30 → Visit 31 | 62 days | ± 14 days |

<sup>&</sup>lt;sup>1</sup>Whenever possible the investigator should arrange study visits within this interval.

Table 2 Intervals between study visits for the investigational vaccine group: Adu1Fx

| Interval | Optimal length of interval <sup>1</sup> | Allowed interval <sup>2</sup> |
|---|---|---|
| Visit 1 (Screening) → Visit 2 (1st vaccination) | 0 to 90 days | - |
| Visit 2 → Visit 7 (2 <sup>nd</sup> vaccination) | 196 days | ± 14 days |
| Visit 7 → Visit 9 | 7 days | ± 1 day |
| Visit 7 → Visit 10 | 30 days | ± 7 days |
| Visit 7 → Visit 11 (Challenge) | 90 days | + 14 days |
| Visit 11 → Visit 30 | 28 days | $\pm$ 7 days |
| Visit 30 → Visit 31 | 62 days | $\pm$ 14 days |

<sup>&</sup>lt;sup>1</sup> Whenever possible the investigator should arrange study visits within this interval.

Table 3 Intervals between study visits for the infectivity control group

| Interval | Optimal length of interval <sup>1</sup> | Allowed interval <sup>2</sup> |
|---|---|---|
| Visit 1b (Screening) → Visit 11 (Challenge) | 0 to 56 days | - |
| Visit 11 → Visit 30 | 28 days | ± 7 days |

<sup>&</sup>lt;sup>1</sup>Whenever possible the investigator should arrange study visits within this interval.

<sup>&</sup>lt;sup>2</sup> Subjects may not be eligible for inclusion in the according-to-protocol (ATP) cohort for analysis of immunogenicity and efficacy if they make the study visit outside this interval.

<sup>&</sup>lt;sup>2</sup> Subjects may not be eligible for inclusion in the ATP cohort for analysis of immunogenicity and efficacy if they make the study visit outside this interval.

<sup>&</sup>lt;sup>2</sup> Subjects may not be eligible for inclusion in the ATP cohort for analysis of immunogenicity and efficacy if they make the study visit outside this interval.

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

The following group names will be used for the statistical analyses:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | AduFx | RTS,S/AS01 <sub>B</sub> full dose administered at Month 0, Month 1 and RTS,S/AS01 <sub>B</sub> 1/5 <sup>th</sup> dose administered at Month 7 |
| 2 | 2PedFx | RTS,S/AS01 <sub>E</sub> double dose administered at Month 0, Month 1 and double dose RTS,S/AS01 <sub>E</sub> 1/5 <sup>th</sup> dose administered at Month 7 |
| 3 | PedFx | RTS,S/AS01 <sub>E</sub> full dose administered at Month 0, Month 1 and RTS,S/AS01 <sub>E</sub> 1/5 <sup>th</sup> dose administered at Month 7 |
| 4 | Adu2Fx | RTS,S/AS01 $_{\rm B}$ full dose at Month 0 and RTS,S/AS01 $_{\rm B}$ 1/5 $^{\rm th}$ dose administered at Month 1, Month 7 |
| 4 | Adu1Fx | RTS,S/AS01 <sub>B</sub> full dose at Month 0 and RTS,S/AS01 <sub>B</sub> 1/5 <sup>th</sup> dose administered at Month 7 |
| 5 | Control | Subjects will not receive any immunization but will undergo sporozoite challenge |

# Two defined pooled groups:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | Р | All subjects who have not been infected by <i>P. falciparum</i> parasitemia (defined by a positive blood slide) during the challenge and were part of one of the vaccinated groups |
| 2 | NP | All subjects who have been infected by <i>P. falciparum</i> parasitemia (defined by a positive blood slide) during the challenge and were part of one of the vaccinated groups |

# 3. OBJECTIVES

# 3.1. Primary objective

# 3.1.1. Efficacy

• To assess the vaccine efficacy against the occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) for each vaccination schedule (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx) versus the infectivity controls.

Refer to Section 4.1 for the definition of the primary endpoint.

# 3.2. Secondary objectives

# 3.2.1. Efficacy

- To assess the time to onset of *P. falciparum* parasitemia (defined by a positive blood slide) for each vaccination schedule (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx) versus the infectivity controls.
- To assess the occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) after vaccine administration for alternative vaccination schedules (2PedFx, PedFx, Adu2Fx, and Adu1Fx) versus the immunization schedule of reference (AduFx).
- To assess the time to onset of *P. falciparum* parasitemia (defined by a positive blood slide) after vaccine administration for alternative vaccination schedules (2PedFx, PedFx, Adu2Fx, and Adu1Fx) versus the immunization schedule of reference (AduFx).

# 3.2.2. Immunogenicity

For each vaccination schedule:

- To evaluate anti-CS repeat region antibody response at specified timepoints.
- To evaluate anti-HBs immunoglobulin G (IgG) antibody response at specified timepoints.

#### 3.2.3. Safety

For each vaccination schedule:

• To assess the safety (unsolicited AEs/AEs of specific interest/serious adverse events [SAEs]) and reactogenicity (solicited AEs).

Refer to Section 4.2 for the definition of the secondary endpoints.

# 3.3. Tertiary objectives

# 3.3.1. Immunogenicity

For each vaccination schedule:

- To evaluate anti-CS repeat region IgG avidity index at specified timepoints.
- To evaluate anti-full length CS protein IgG concentrations and anti-C terminal portion of the protein (C-term) IgG concentrations at specified timepoints.
- To evaluate anti-full length CS protein and anti-C-term IgG avidity at specified timepoints.

Note: other immuno-assays evaluating the immune response targeting the CS and HBsAg might be performed.

Refer to Section 4.3 for the definition of the tertiary endpoints.

#### 4. ENDPOINTS

# 4.1. Primary endpoint

# 4.1.1. Efficacy

- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>B</sub> administered as full doses at Month 0 and Month 1 and 1/5<sup>th</sup> dose at Month 7 (AduFx group) versus infectivity controls.
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>E</sub> administered as double dose at Month 0 and Month 1 and double 1/5<sup>th</sup> dose at Month 7 (2PedFx group) versus infectivity controls.
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>E</sub> administered as full doses at Month 0 and Month 1 and 1/5<sup>th</sup> dose at Month 7 (PedFx group) versus infectivity controls.
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>B</sub> administered as one full dose at Month 0 and 1/5<sup>th</sup> doses at Month 1 and Month 7 (Adu2Fx group) versus infectivity controls.
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>B</sub> administered as one full dose at Month 0 and 1/5<sup>th</sup> doses at Month 7 (Adu1Fx group) versus infectivity controls.

# 4.2. Secondary endpoints

# 4.2.1. Efficacy

- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>E</sub> administered as double dose at Month 0 and Month 1 and double 1/5<sup>th</sup> dose at Month 7 (2PedFx group) versus immunization schedule of reference (AduFx group).
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>E</sub> administered as full doses at Month 0 and Month 1 and 1/5<sup>th</sup> dose at Month 7 (PedFx) versus immunization schedule of reference (AduFx group).
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>B</sub> administered as one full dose at Month 0 and 1/5<sup>th</sup> full dose at Month 1 and Month 7 (Adu2Fx) versus immunization schedule of reference (AduFx group).
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>B</sub> administered as one full dose at Month 0 and 1/5<sup>th</sup> full doses at Month 7 (Adu1Fx) versus immunization schedule of reference (AduFx group).
- Time to onset of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge in each vaccination schedule versus immunization schedule of reference (AduFx group).
- Time to onset of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge in each vaccination schedule versus infectivity controls.

# 4.2.2. Immunogenicity

- For each vaccination schedule, the immune response to the CS antigen of the investigational vaccine:
  - Anti-CS repeat region antibody concentrations before vaccine administration (Day 0), one month post-Dose 2 (Day 58), six months post-Dose 2 (Day 196), one month post-Dose 3 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx groups and before vaccine administration (Day 0), before Dose 2 (Day 196), one month post-Dose 2 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from Adu1Fx group.

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

- For each vaccination schedule, the immune response to the hepatitis B antigen of the investigational vaccine:
  - Anti-HBs IgG antibody concentrations before vaccine administration (Day 0), one month post-Dose 2 (Day 58), six months post-Dose 2 (Day 196), one month post-Dose 3 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx groups and before vaccine administration (Day 0), before Dose 2 (Day 196), one month post-Dose 2 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from Adu1Fx group.

# 4.2.3. Safety

- Safety and reactogenicity of the investigational vaccine for each vaccination schedule:
  - Occurrence of solicited local and general AEs within seven days (day of vaccination and six subsequent days) after each vaccination.
  - Occurrence of unsolicited AEs within 30 days (day of vaccination and 29 subsequent days) after each vaccination, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification.
  - Occurrence of AEs within 30 days (day of challenge and 29 subsequent days) after challenge, according to the MedDRA classification.
  - Occurrence of SAEs (all, fatal, related to investigational vaccine) within 30 days (day of vaccination and 29 subsequent days) after each vaccination, according to the MedDRA classification.
  - Occurrence of SAEs (all, fatal, related to investigational vaccine) during the whole study period (from Dose 1 [Day 0] up to study conclusion [Day 376]), according to the MedDRA classification.
  - Occurrence of AEs and SAEs leading to withdrawal from further vaccination from Dose 1 (Day 0) up to study conclusion (Day 376), according to the MedDRA classification, for each vaccinated subject.
  - Occurrence of pIMDs from Dose 1 (Day 0) up to study conclusion (Day 376),
     according to the MedDRA classification, for each vaccinated subject.
  - Occurrence of meningitis from Dose 1 (Day 0) up to study conclusion (Day 376), according to the MedDRA classification, for each vaccinated subject.
  - Occurrence of abnormal laboratory values at screening, Day 35, Day 58, Day 203, Day 226, the day of first parasitemia, and Day 314 for each vaccinated subject and at screening, the day of first parasitemia and Day 314 for the infectivity control subjects.

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

- Safety after sporozoite challenge in the infectivity control group.
  - Occurrence of AEs within 30 days (day of challenge and 29 subsequent days) after challenge, according to the MedDRA classification.
  - Occurrence of SAEs (all, fatal, related) from day of challenge (Day 286) to the end of the challenge phase (Day 314), according to the MedDRA classification.

# 4.3. Tertiary endpoints

# 4.3.1. Immunogenicity

- For each vaccination schedule, the immune response to the CS antigen of the investigational vaccine:
  - Anti-CS repeat region IgG avidity index before vaccine administration (Day 0), one month post-Dose 2 (Day 58), six months post-Dose 2 (Day 196), one month post-Dose 3 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx groups and before vaccine administration (Day 0), before Dose 2 (Day 196), one month post-Dose 2 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from Adu1Fx group.
  - Anti-full length CS protein IgG concentrations and anti-C-term IgG concentrations before vaccine administration (Day 0), one month post-Dose 2 (Day 58), six months post-Dose 2 (Day 196), one month post-Dose 3 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx groups and before vaccine administration (Day 0), before Dose 2 (Day 196), one month post-Dose 2 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from Adu1Fx group.
  - Anti-full length CS protein and anti-C-term IgG avidity before vaccine administration (Day 0), one month post-Dose 2 (Day 58), six months post-Dose 2 (Day 196), one month post-Dose 3 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx groups and before vaccine administration (Day 0), before Dose 2 (Day 196), one month post-Dose 2 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from Adu1Fx group.

Note: other immuno-assays evaluating the immune response targeting the CS and HBsAg might be performed.

# 5. ANALYSIS SETS

#### 5.1. Definition

Note that in order to align to ICH and CDISC terminology the According To Protocol (ATP) cohort has been renamed the Per-Protocol Set (PPS).

#### 5.1.1. Enrolled Set

The Enrolled Set will include all screened subjects who provide informed consent and provide demographic and/or other baseline screening measurements, regardless of the subject's randomization and vaccination status in the trial, and receive a subject ID.

# 5.1.2. Intent-to-treat set (ITTS)

The Intent-To-Treat Set (ITTS) will include all subjects who received at least one dose of study vaccine. The ITTS analysis will be performed per treatment actually administered. All challenged infectivity controls will also be included and will be presented as a separate study group.

# 5.1.3. Solicited Safety Set

The solicited Safety Set will include all subjects who received at least one dose of study vaccine and had solicited safety data.

# 5.1.4. Per-Protocol Set for analysis of immunogenicity and efficacy (PPS for analysis of immunogenicity and efficacy)

The PPS for analysis of immunogenicity and efficacy will include all subjects included in the ITTS who fulfilled all eligibility criteria and received all vaccinations according to protocol procedures within the protocol specified intervals, did not use any medication, vaccine or blood products forbidden by the protocol, did not report any underlying medical condition influencing the efficacy response, had available data concerning immunogenicity endpoint measures, and underwent *P. falciparum* challenge. This will include subjects for whom assay results are available for antibodies against at least one study vaccine antigen after vaccination.

# 5.1.5. Adapted Per-Protocol Set for analysis of efficacy (Adapted PPS for analysis of efficacy)

The Adapted PPS for analysis of efficacy will include all subjects included in the ITTS who fulfilled all eligibility criteria and received all vaccinations according to protocol procedures within the protocol specified intervals and underwent *P. falciparum* challenge.

Statistical Analysis Plan Amendment 1 Final

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

#### 5.2.1. Elimination from ITTS

Code 1030 (Study vaccine not administered at all) for all subjects except those from the infectivity control group and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ITTS.

### 5.2.2. Elimination from the Solicited Safety Set

Code 1030 (study vaccine not administered at all), code 900 (invalid informed consent or fraud data) and code 1160 (no post-vaccination solicited safety data) will be used for identifying subjects eliminated from the solicited safety set.

# 5.2.3. Elimination from the PPS for analysis of immunogenicity and efficacy

#### 5.2.3.1. Excluded subjects

A subject will be excluded from the PPS analysis of immunogenicity and efficacy analysis under the following conditions

| Code | Condition under which the code is used |
|---|---|
| 900 | Invalid informed consent or fraud data |
| 1030 | Study vaccine not administered at all |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol |
| | Any investigational or non-registered vaccine other than the study vaccines used during the study period. |
| | • A vaccine not foreseen by the study protocol administered during the period starting seven days before each dose and ending seven days after each dose of vaccines administration. |
| 1070 | Vaccination not according to protocol |
| | Incomplete vaccination course before treatment withdrawal or subject study conclusion. |
| | • Administration not according to protocol for reason specified by the investigator, other than side, site and route. |
| | Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number). |
| | Study vaccine RTS,S/AS01 not prepared as per protocol |

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

| Code | Condition under which the code is used |
|---|---|
| 1080 | Good Manufacturing Practice No-Go: Vaccine temperature deviation |
| 1090 | Expired vaccine administered |
| 2010 | Protocol violation (inclusion/exclusion criteria) |
| | Eligibility criteria not met with an impact on immunogenicity data |
| 2040 | Administration of any medication forbidden by the protocol which may influence the efficacy endpoints |
| | Any investigational or non-registered product drug other than the study vaccines used during the study period. |
| | • Immunosuppressants or other immune-modifying drugs administered chronically (i.e. more than 14 days in total) during the study period. For corticosteroids, this will mean prednisone ≥ 20 mg/day (for adult subjects), or equivalent. Inhaled and topical steroids are allowed. |
| | • Long-acting immune-modifying drugs administered at any time during the study period (e.g. infliximab). |
| | Immunoglobulins and/or any blood products administered during the study period. |
| | • Drugs known to have anti- <i>Plasmodium</i> properties, used during the challenge period before identification of parasitemia. |
| 2050 | Underlying medical condition forbidden by the protocol which may influence the efficacy endpoints |
| 2080 | Subjects did not comply with vaccination schedule |
| | (See Table 1, Table 2, Table 3) |
| 2090 | Subjects did not comply with blood sampling schedule |
| | (See Table 1, Table 2, Table 3) |
| 2100 | Serological results not available for anti-CS at all post-vaccination visits |
| 2120 | Obvious incoherence or abnormality or error in immunogenicity (antibody) data |
| 3000 | Subject did not undergo challenge |

Statistical Analysis Plan Amendment 1 Final

# 5.2.4. Elimination from the Adapted PPS for analysis of efficacy

# 5.2.4.1. Excluded subjects

A subject will be excluded from the Adapted PPS analysis of efficacy analysis under the following conditions:

| Code | Condition under which the code is used |
|---|---|
| 900 | Invalid informed consent or fraud data |
| 1030 | Study vaccine not administered at all |
| 1070 | Vaccination not according to protocol |
| | Incomplete vaccination course before treatment withdrawal or subject study conclusion. |
| | Administration not according to protocol for reason specified by the investigator, other than side, site and route. |
| | Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number). |
| | Study vaccine RTS,S/AS01 not prepared as per protocol |
| 3000 | Subject did not undergo challenge |

# 5.3. Important protocol deviations not leading to elimination from per-protocol analysis set

Important protocol deviations not leading to elimination from PPS are defined in MALARIA-092 (205081) Protocol Deviation Management Plan.

PPD

(MALARIA-092 (205081) Protocol Deviation Management Plan)

#### 6. STATISTICAL ANALYSES

Note that standard data derivation rules and statistical methods are described in Annex 1 and will not be repeated below.

# 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

A study flow table (consort) will be generated to present the number of subjects screened, randomized, receiving doses and included in the PPS for analyses.

The analysis of demographics will be performed on the ITTS and on the PPS for analysis of immunogenicity and efficacy.

Demographic characteristics (age at first vaccination in years for the vaccinated groups and at the time of the screening for the control group, gender, and race) will be summarized by group and overall using descriptive statistics:

- Frequency tables will be generated for categorical variables such as race.
- Mean, median, standard deviation (SD) and range will be provided for continuous data such as age.
  - Withdrawal status will be summarized by group using descriptive statistics:
- The number of subjects enrolled into the study as well as the number of subjects excluded from PPS for analyses will be tabulated.
- The number of withdrawn subjects will be tabulated according to the reason for withdrawal.

# 6.2. Exposure

#### 6.2.1. Analysis of exposure planned in the protocol

The number and percentages of subjects with vaccination will be summarized overall and by group for all groups where a vaccination is part of the study procedure. The analysis of exposure will be performed on the ITTS.

# 6.3. Efficacy analysis

# 6.3.1. Analysis of efficacy planned in the protocol

The analysis of efficacy will be performed on the PPS for analysis of immunogenicity and efficacy.

Efficacy will be assessed by comparison of *P. falciparum* parasitemia incidence and time to onset of *P. falciparum* parasitemia after sporozoite challenge.

Vaccine efficacy (VE) is defined as 100\*(1-Relative Risk). Relative risk of infection and 95% CI will be calculated.

Fisher's Exact test will be used for the comparison of *P. falciparum* parasitemia incidence after challenge between each one of the vaccine groups (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx) and the infectivity control group.

Kaplan-Meier analysis will be performed on time to onset of *P. falciparum* parasitemia, for comparisons between each one of the vaccine groups (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx) and the infectivity control group, using the log-rank statistic.

The same methodology will be applied for the evaluation of the vaccinated groups versus the immunization schedule of reference (AduFx group).

All statistical tests will be two-tailed at 5% significance level.

#### 6.3.2. Additional considerations

#### 6.3.2.1. Case definition

The primary case definition of P. falciparum infection is an asexual blood stage P. falciparum parasite density > 0 detected by blood slide reading.

# 6.3.2.2. Risk periods

For the analyses of time to onset of parasitemia (Kaplan-Meier and Log-Rank), time at risk will start on first day of challenge. Time at risk will be censored on protocol visit D314 (28 days post challenge), drop-out date, start date of antimalarial treatment or date meeting an endpoint, whichever occurs first. Time at risk will be calculated as: censor date – date challenge + 1.

For the analysis of proportion affected (relative risk), all subjects included in the PPS for analysis of immunogenicity and efficacy will be considered at risk of infection and no censoring or elimination will be applied for subjects not completing the entire protocol defined post challenge follow-up (visit D314 - 28 days post challenge).

# 6.4. Immunogenicity analysis

# 6.4.1. Analysis of immunogenicity planned in the protocol

The analysis of immunogenicity will be performed on the PPS for analysis of immunogenicity and efficacy.

For each study group, at each timepoint that a blood sample result is available:

The percentage of subjects with seropositive levels of anti-CS (proportion of subjects with anti-CS antibody concentrations  $\geq$  1.9 EU/ml) with 95% CI will be determined at specified blood sampling timepoints in each group (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx). Anti-CS antibody concentrations will be summarized by GMC. Anti-CS antibody concentrations will be displayed using reverse cumulative curves. Similar analysis will be performed for the anti-full length CS protein (proportion of subjects with anti-CS antibody titres  $\geq$  200 1/DIL) and anti-C-term antibodies (proportion of subjects with anti-CS antibody concentrations  $\geq$ 100 EPT).

The percentage of subjects with seroprotection levels of anti-HBs (anti-HBs antibody concentrations ≥ 10 mIU/ml) with 95% CI will be determined at specified blood sampling timepoints in each group (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx). Anti-HBs antibody concentrations will be summarized by GMC. Anti-HBs antibody concentrations will be displayed using reverse cumulative curves.

Anti-CS, anti-full length CS protein and anti-CS avidity index will be summarized by mean, SD, median and quartile and box and whiskers plots will be generated.

#### 6.4.2. Additional considerations

In addition to the previous analyses, the immunogenicity analyses will be performed per protection status (P and NP) overall (pooled vaccine groups) and within each vaccine group.

A comparisons of the log-transformed means of anti-CS antibodies (repeated, full length, C-Term and avidity index) post vaccination and at the time of the challenge and for P vs NP (Student 2-Sample Test) will be performed.

Exploratory analyses using logistic regression models will be evaluated to describe the relationship between immune read outs and the probability of infection (P vs NP). Explanatory variables will include all or a part of available immune read outs at time of analysis (anti-CS, anti-full length CS protein, avidity index).

In a first step, immune responses will be plotted by group and protection status as well as cross-tabulated to understand potential correlation structures. Then, relevant models will be constructed to evaluate what are the independent predictors of protection, both pooled over the treatment groups (is/are there a generic driver(s)?) and by treatment schedule/including interactions (is protection mediated through different mechanisms between schedules?).

# 6.5. Analysis of safety

# 6.5.1. Analysis of safety planned in the protocol

The analysis of safety will be performed on the ITTS.

The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period after each vaccine dose and overall will be tabulated with exact 95% CI. The percentage of doses followed by at least one local AE (solicited and unsolicited), by at least one general AE (solicited and unsolicited) and by any AE during the 7-day or 30-day follow-up period will be tabulated with exact 95% CI. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination and for any Grade 3 AEs considered related to vaccination.

The percentage of subjects reporting each individual solicited local AE (any grade and Grade 3) and each individual solicited general AE (any grade, Grade 3, any related, Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period (Day 0-6) after each vaccine dose and overall will be tabulated for each group. Similarly, the percentage of doses followed by each individual solicited local and general AE will be tabulated, for the overall and for each vaccination course, with exact 95% CI.

For fever (fever is defined as temperature  $\geq 37.5^{\circ}\text{C}/99.5^{\circ}\text{F}$  for oral, axillary or tympanic route, or  $\geq 38.0^{\circ}\text{C}/100.4^{\circ}\text{F}$  for rectal route), the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the first seven days (Day 0-6) after each vaccine dose and overall will be tabulated. Similar tabulations will be performed for any fever with a causal relationship to vaccination and Grade 3 (> 39.0°C) causally related fever. The maximum temperature reported over the 7-day follow-up period (Day 0-6) overall doses will be tabulated.

The percentage of subjects reporting unsolicited AEs within 30 days (Day 0-29) after each vaccine dose (overall doses) and percentage of subjects reporting AEs after the sporozoite challenge will be tabulated by group and by MedDRA preferred term with exact 95% CI. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs and for Grade 3 causally related unsolicited AEs.

The percentage of subjects reporting SAEs (all, fatal, related) occurring within 30 days (day of vaccination and 29 subsequent days) after each dose of study vaccine, classified by the MedDRA preferred term level will be tabulated with exact 95% CI.

The percentage of subjects reporting SAEs (all, fatal, related) occurring from Dose 1 (Day 0) until last study visit (Day 376), classified by the MedDRA preferred term level will be tabulated with exact 95% CI.

The percentage of subjects reporting SAEs (all, fatal, related) occurring from day of challenge (Day 286) to the end of the challenge phase (Day 314), according to the MedDRA classification will be tabulated with exact 95% CI.

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

Subjects reporting pregnancies will be described.

The percentage of subjects reporting an AE or SAE leading to withdrawal from further vaccination from Dose 1 (Day 0) until last study visit (Day 376), classified by MedDRA preferred term level, will be tabulated with exact 95% CI.

The percentage of vaccinated subjects reporting AEs of specific interest (meningitis and pIMDs) from Dose 1 (Day 0) until last study visit (Day 376), classified by MedDRA preferred term level, will be tabulated with exact 95% CI.

Biochemistry (ALT, AST and creatinine) and hematological (hemoglobin, WBC and platelets) laboratory values will be presented by visit according to toxicity grading scales and tabulated by group.

The normal ranges and toxicity grading for laboratory safety parameters used in this study are presented in Table 4

Table 4 Toxicity grading scales for blood testing

| Adverse event | Intensity grade | Intensity* |
|---|---|---|
| Hemoglobin (males) | Normal range | ≥12.5 g/dl |
| | 1 | < 12.5 but ≥ 11.0 g/dl |
| | 2 | < 11.0 but ≥ 10.0 g/dl |
| | 3 | < 10.0 g/dl |
| Hemoglobin (females) | Normal range | ≥11.5 g/dl |
| | 1 | < 11.5 but ≥ 10.5 g/dl |
| | 2 | < 10.5 but ≥ 9.5 g/dl |
| | 3 | < 9.5 g/dl |
| Increase in leukocytes | Normal range | ≤10799 cells/mm <sup>3</sup> |
| (WBC) | 1 | 10800 - 15000 cells/mm <sup>3</sup> |
| , | 2 | 15001 - 20000 cells/mm <sup>3</sup> |
| | 3 | > 20001 cells/mm <sup>3</sup> |
| Decrease in leukocytes | Normal range | ≥3200 cells/mm <sup>3</sup> |
| (WBC) | 1 | 2500 - 3199 cells/mm <sup>3</sup> |
| | 2 | 1500 - 2499 cells/mm <sup>3</sup> |
| | 3 | < 1500 cells/mm <sup>3</sup> |
| Decrease in platelets | Normal | ≥140000 cells/mm <sup>3</sup> |
| | 1 | 125000 - 139000 cells/mm <sup>3</sup> |
| | 2 | 100000 - 124000 cells/mm <sup>3</sup> |
| | 3 | < 100000 cells/mm <sup>3</sup> |
| Alanine Aminotransferase | Normal range | Below ULN (60 U/I for males; 40 U/I for females) |
| | 1 | 1.1 - 2.5 x ULN |
| | 2 | 2.6 – 5 x ULN |
| | 3 | > 5 x ULN |
| Aspartate Aminotransferase | Normal range | Below ULN (40 U/I for males; 35 U/I for females) |
| | 1 | 1.1 - 2.5 x ULN |
| | 2 | 2.6 – 5 x ULN |
| | 3 | > 5 x ULN |
| Creatinine (males) | Normal range | ≤1.39 mg/dl |
| | 1 | 1.4 - 1.79 mg/dl |
| | 2 | 1.8 - 2.0 mg/dl |
| | 3 | > 2.0 mg/dl |
| Creatinine (females) | Normal range | ≤1.29 mg/dl |
| | 1 | 1.3 – 1.69 mg/dl |
| | 2 | 1.7 – 1.9 mg/dl |
| | 3 | >1.9 mg/dl |

ULN: upper limit of normal range

The percentage of subjects using concomitant medication (any medication, any antipyretic and any prophylactic medication, respectively) during the 7-day follow-up period (Day 0-6) after vaccination will be summarized by group after each dose and overall. The percentage of subjects using concomitant medication during the entire sporozoite challenge (D286-314) will be summarized by group.

<sup>\*</sup> Grading scale adapted from [FDA guidance for industry toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (September 2007)].

Statistical Analysis Plan Amendment 1 Final

#### 6.5.2. Additional considerations

A summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes:

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| FATIGUE | 10016256 | Fatigue |
| FEVER | 10016558 | Fever |
| GASTROINTESTINAL | 10017944 | Gastrointestinal disorder |
| HEADACHE | 10019211 | Headache |
| PAIN | 10022086 | Injection site pain |
| REDNESS | 10022098 | Redness at injection site |
| SWELLING | 10053425 | Swelling at injection site |

The following analysis will be performed if at least 5 subjects have used concomitant vaccination during the 7-day follow-up period (Day 0-6) after study vaccination during the full study period.

The percentage of subjects using any concomitant vaccination during the 7-day follow-up period (Day 0-6) after study vaccination will be summarized by group after each dose and overall. The percentage of subjects using concomitant vaccination during the entire sporozoite challenge will be summarized by group.

Note that the study will be converted in CDISC. Accordingly protocol Day 0-Day N will be replaced by Day 1-Day N+1 for the statistical analysis.

# 7. ANALYSIS INTERPRETATION

All the analyses performed during this study will be descriptive.

### 8. CONDUCT OF ANALYSES

# 8.1. Sequence of analyses

The analyses will be performed stepwise:

- An interim analysis to allow an internal decision for the choice of the booster dose in study Malaria-102 will be performed as soon as the results of the challenge phase will be available on data as clean as possible. This analysis will be descriptive and performed on the Adapted PPS for analysis of efficacy.
- When all the remaining data up to Day 376 will be available, the main analysis will be performed. An integrated study report will be written.

# 8.2. Statistical considerations for interim analyses

A descriptive analysis to evaluate VE against infection of *P. falciparum* will be performed on the Adapted PPS for analysis of efficacy at the time of the interim analysis. Note that the main objective of the study linked to this endpoint will be analysed at the end of the study, on the PPS for analysis of immunogenicity and efficacy and can output different results.

### 9. CHANGES FROM PLANNED ANALYSES

The Total vaccinated cohort (TVC) defined in the protocol has been replaced by the Intent-To-Treat Set (ITTS) to include both subjects vaccinated and subjects from the infectivity control group in the same cohort.

An interim analysis has been added to allow an internal decision for the choice of the booster dose in study Malaria-102. This analysis will be descriptive and performed on data as cleaned as possible.

To allow an interim analysis as close as possible to the main analysis, an Adapted PPS for analysis of efficacy has been created.

An analysis of concomitant vaccination has been added to assess any effect on immune response or safety.

A Solicited Safety Set has been added in the analysis set section to fit with the new statistical rules and layouts applicable from the 12<sup>th</sup> of November.

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS, Annex). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulations of individual data such as listings of SAEs. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

Statistical Analysis Plan Amendment 1 Final

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day & month are missing, 30 June is used.
- Onset day for an event (AE, medication, vaccination): The onset day is the number of days between the last study vaccination & the onset/start date of the event. This is 1 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.
- Duration: Duration of an event is expressed in days. It is the number of days between the start & the stop dates + 1. Therefore duration is 1 day for an event starting & ending on the same day.

#### 11.2.2. Dose number

- The study dose number is defined in reference to the number of study visits at which vaccination occurred. More specifically dose 1 refers to all vaccines administered at the first vaccination visit while dose 2 corresponds to all vaccinations administered at the second vaccination visit even if this is the first time a product is administered to the subject.
- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an AE begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose. In case a study dose is not administered (eg dose 2) and an event occurs after the subsequent study dose (eg 3rd study dose), the relative dose of the event will be study dose associated to the subsequent study dose (eg dose 3).
- The number of doses for a product is the number of times the product was administered to a subject.
- The incidence per dose is the number of vaccination visits at which an event was reported among all vaccination visits.

### 11.2.3. Demography

- Age: Age at the reference activity, computed as the number of years between the date of birth and the reference activity. Note that due to incomplete date, the derived age may be incorrect by 1 year when month is missing from the birthdate. This may lead to an apparent inconsistency between the derived age and the eligibility criteria/the age category used for randomization.
- Conversion of weight to kg

The following conversion rule is used:

Weight in Kilogrammes= weight in Pounds / 2.2 + weight in Ounces / 35.2

The result is rounded to 2 decimals.

• Conversion of height to cm

The following conversion rule is used:

Height in Centimetres = Height in Feet \* 30.48 + Height in Inches \* 2.54

The result is rounded to the unit (ie no decimal).

Conversion of temperature to °C

The following conversion rule is used:

- Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

# 11.2.4. Immunogenicity

- For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.
- The Geometric Mean Concentrations (GMCs) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMC calculation. The cut-off value is defined by the laboratory before the analysis.
- The percentage of subjects seropositive/seroprotected and associated two-sided 95% Clopper-Pearson confidence intervals (CIs) will be computed by vaccine group for each available immunogenicity monitoring.
- A subject seropositive for anti-CS antibody will be a subject whose antibody concentration will be greater than or equal to the cut-off value (anti-CS ≥ 1.9 EU/ml).
- Seroprotection rate for anti-HBs antibody is defined as the percentage of subjects with antibody concentration greater than or equal to an established cut-off (anti-HBs ≥ 10 mIU/ml).

### 11.2.5. Safety

- Handling of missing data: subjects who missed reporting symptoms (unsolicited or concomitant medications) will be treated as subjects without symptoms (unsolicited or concomitant medications, respectively). In case of significant non-compliance of study procedures for reporting symptoms, the analysis plan will be reassessed to ensure more accurate reporting of study data by further analysis.
- For the analysis of solicited symptoms, missing or non-evaluable measurements will
  not be replaced. Therefore the analysis of the solicited symptoms based on the ES
  will include only subjects/doses with documented safety data (i.e. symptom
  screen/sheet completed).
- For a given subject and the analysis of solicited symptoms within 7 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the ES will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed). More specifically the following rules will be used:
  - Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
  - Subjects who documented the presence of a solicited symptom and fully or
    partially recorded daily measurement over the solicited period will be included
    in the summaries at that dose and classified according to their maximum
    observed daily recording over the solicited period.
  - Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be assigned to the lowest intensity category at that dose (i.e., 37.5°C for fever or grade 1 for other symptoms).
  - Doses without symptom sheets documented will be excluded.
- For analysis of unsolicited AEs, such as SAEs or AEs by primary MedDRA term, and for the analysis of concomitant medications, all vaccinated subjects will be considered.
- For the analysis, temperatures will be coded as follows:

| Grade | Temperature |
|-------|--------------------------------------------|
| 0 | < 37.5°C (< 99.5°F) |
| 1 | ≥ 37.5°C (≥ 99.5°F) to ≤ 38.0°C (100.4°F) |
| 2 | > 38.0°C (> 100.4°F) to ≤ 39.0°C (102.1°F) |
| 3 | > 39.0°C (102.1°F) |

• For the analysis, local injection site redness and swelling will be coded as follows:

| Grade | Temperature |
|-------|---------------------|
| 0 | 0 mm |
| 1 | > 0 to ≤ 50 mm |
| 2 | > 50 mm to ≤ 100 mm |
| 3 | > 100 mm |

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for | N used for deriving % per dose for |
|---|---|---|
| Event | Vaccination phase | Vaccination phase |
| Concomitant | All subjects with study vaccine | All study visits with study vaccine |
| vaccination | administered | administered |
| Solicited general | All subjects with at least one solicited | All study visits with study vaccine |
| symptom | general symptom documented as either | administered and with at least one solicited |
| | present or absent (i.e., symptom screen | general symptom documented as either |
| | completed) | present or absent (i.e., symptom screen |
| | | completed) |
| Solicited local | All subjects with at least one solicited local | All study visits with study vaccine |
| symptom | symptom documented as either present or | administered and with at least one solicited |
| | absent (i.e., symptom screen completed) | local symptom documented as either |
| | | present or absent (i.e., symptom screen |
| | | completed) |
| Unsolicited symptom | All subjects with study vaccine | All study visits with study vaccine |
| | administered | administered |
| Concomitant | All subjects with study vaccine | All study visits with study vaccine |
| medication | administered | administered |

• Related dose: The related dose for an event (e.g., AE, medication, vaccination,...) is the study dose given before an event. In case the event takes place on a day a study dose is given, if the investigator has indicated the timing (before or after the vaccination) the related dose for this event is the most recent study dose given before this event. If the investigator has not indicated the timing, the related dose will be that of the study dose even if the event actually took place before.

#### Number of decimals displayed:

The following decimal description from the decision rules will be used for demography, efficacy, immunogenicity and safety/reactogenicity results.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| Demographic characteristics | Mean, median age | 1 |
| Demographic characteristics | SD (age) | 1 |
| Reactogenicity | Mean, Min, Q1, Median, Q3, Max for duration | 1 |
| All summaries | p-value | 3 |

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 subjects in each tabulated group
- one decimal when there are at least 50 subjects in at least one tabulated group
  - Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

- The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.
- Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

# **Differences in percentages**

Differences in percentages and their corresponding confidence limits will be displayed with one more decimal than the maximum number used to display the individual percentages, for example the difference between two percentages displayed with one decimal will be displayed with two decimals.

#### Serological summary statistics

The number of decimals used when displaying geometric mean titers (GMT) or concentrations (GMC) and their confidence limits is shown in the following table:

| GMT or GMC value | Number of decimals to display |
|------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT or GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). For example, if GMT or GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.
205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

#### **12**. **ANNEX 2: TABLES, FIGURES AND LISTINGS**

#### 12.1. **Demographics & baseline characteristics**

| Template # | Table Title | Output destination | Template name |
|---|---|---|---|
| Template 1 | Summary of subject disposition from Enrolled Set to Randomized/Intent-To-Treat Set (Enrolled set) | Post-text | TCONSORT1PART1/Specific |
| Template 2 | Summary of subject disposition from Intent-To-<br>Treat Set to Per Protocol Set for analysis of<br>immunogenicity and efficacy (Intent-to-treat set) | Post-text / in-text | TCONSORT1PART3 |
| Template 3 | Summary of visit attendance (Intent-to treat set) | Post-text | TMH1SOCPT |
| Template 3 | Summary of visit attendance (Per protocol set for analysis of immunogenicity and efficacy for efficacy) | Post-text | TMH1SOCPT |
| Template 4 | Summary of study completion with reasons for withdrawal (Intent-to-treat set) | Post-text / Web disclosure | TSL1WITHDRAWAL |
| Template 4 | Summary of study completion with reasons for withdrawal (Per protocol set for analysis of immunogenicity and efficacy for efficacy) | Post-text | TSL1WITHDRAWAL |
| Template 5 | Summary of important protocol deviations leading to elimination (Intent-to-treat set) | In-text / Post-text | TDV1PROTDEV |
| Template 6 | Deviations from protocol for age and intervals between study visits (Intent-to-treat set) | Post-text | TDEVINT1INTVAL |
| Template 6 | Deviations from protocol for age and intervals<br>between study visits (Per protocol set for<br>analysis of immunogenicity and efficacy for<br>efficacy) | Post-text | TDEVINT1INTVAL |
| Template 10 | Exposure to study vaccine (Intent-to-treat set) | In-text / Post-text | TEXOVW1EXPOBYBYVAC |
| Template 7 | Summary of demographic characteristics and baseline characteristics (Intent-to-treat set) | In-text / Post-text | TSL1DEMOG |
| Template 7 | Summary of demographic and baseline characteristics (Per protocol set for analysis of immunogenicity and efficacy for efficacy) | Post-text / in-<br>text/Synopsis | TSL1DEMOG |
| Template 7 | Summary of demographic and baseline characteristics by protection status (Per protocol set for analysis of immunogenicity and efficacy for efficacy) | Post-text | TSL1DEMOG |
| Template 8 | Summary of demographic characteristics and baseline characteristics (Enrolled set) | Web posting | TSL1DEMOG |
| Template 9 | Summary of previous Hepatitis B vaccination (Intent-to-treat set) | Post-text | Specific |
| Template 9 | Summary of previous Hepatitis B vaccination (Per protocol set for analysis of immunogenicity and efficacy for efficacy) | Post-text | Specific |
| Template 32 | Minimum and maximum visit dates (intent-to-treat) | Annex | TACTIV1DATE |

# 12.2. Efficacy

| Template # | Table / Figure Title | Output destination | Template name |
|---|---|---|---|
| Template 11 | Parasitemia incidence defined by a positive blood slide and vaccine efficacy of each vaccination schedule versus Control group during challenge phase (Per protocol set for analysis of immunogenicity and efficacy) | Post-text / in-<br>text / Web<br>disclosure/Syn<br>opsis | Specific |
| Template 12 | Time to onset of parasitemia in each vaccination schedule versus Control (by blood slide) (Per protocol set for analysis of immunogenicity and efficacy) | Post-text / Web disclosure | Specific |
| Template 12 | Time to onset of parasitemia in each vaccination schedule versus AduFx (by blood slide) (Per protocol set for analysis of immunogenicity and efficacy) | Post-text/ Web disclosure | Specific |
| Template 13 | Cumulative incidence of parasitemia onset defined by positive<br>blood slide for all groups (Per protocol set for analysis of<br>immunogenicity and efficacy) | Post-text | Specific |
| Template 11 | Parasitemia incidence defined by a positive blood slide and vaccine efficacy of each vaccination schedule versus AduFx during challenge phase (Per protocol set for analysis of immunogenicity and efficacy) | Post-text/ Web disclosure | Specific |

# 12.3. Immunogenicity

| Template # | Table / Figure Title | Output destination | Template name |
|---|---|---|---|
| Anti-CS antibo | odies (repeat) | | |
| Template 14 | Number and percentage of subjects with anti-CS (repeat) equal or above 1.9 EU/mL and GMCs (Per protocol set for analysis of immunogenicity and efficacy) | Post-text / in-<br>text / Web<br>disclosure/Syno<br>psis | TIS1GMT |
| Template 14 | Number and percentage of subjects with anti-CS (repeat) equal or above 1.9 EU/mL and GMCs by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | TIS1GMT |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (repeat) post-vaccination (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (repeat) post-vaccination by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (repeat) at the time of the challenge (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (repeat) at the time of the challenge by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 17 | Box and whiskers plot of anti-CS antibodies (repeat) at post-<br>vaccination and the day of the challenge (Per protocol set<br>for analysis of immunogenicity and efficacy) | Post-text | Specific |
| Template 17 | Box and whiskers plot of anti-CS antibodies (repeat) at post-<br>vaccination and the day of the challenge by protection status<br>(Per protocol set for analysis of immunogenicity and<br>efficacy) | Post-text | Specific |

| Template # | Table / Figure Title | Output destination | Template name |
|---|---|---|---|
| Template 18 | Evolution over time for anti-CS antibodies (repeat) by group (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | Specific |
| Template 18 | Evolution over time for anti-CS antibodies (repeat) per protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | Specific |
| Template 16 | Comparison of the log-transformed means of the anti-CS (repeat) antibodies at post-vaccination and at the time of the challenge of each vaccination schedule versus AduFx groups (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | specific |
| Template 16 | Comparison of the log-transformed means of the anti-CS (repeat) antibodies at post-vaccination and at the time of the challenge between Protected and Non-Protected groups (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | specific |
| Anti-CS antibo | dies (full length) | • | |
| Tamorla (c. 4.4 | Must be and according of a 12 to 20 of 20 | Deet to 1 | TICACNAT |
| Template 14 | Number and percentage of subjects with anti-CS (full length) equal or above 200 1/DIL and GMTs (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | TIS1GMT |
| Template 14 | Number and percentage of subjects with anti-CS (full length) equal or above 200 1/DIL and GMTs by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | TIS1GMT |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (full length) at post-vaccination (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (full length) at post-vaccination by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (full length) at the time of the challenge (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (full length) at the time of the challenge by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 17 | Box and whiskers plot of anti-CS antibodies (full length) at post-vaccination and the day of the challenge (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | Specific |
| Template 17 | Box and whiskers plot of anti-CS antibodies at post-<br>vaccination and the day of the challenge (full length) by<br>protection status (Per protocol set for analysis of<br>immunogenicity and efficacy) | Post-text | Specific |
| Template 18 | Evolution over time for anti-CS antibodies (full length) by group (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | Specific |
| Template 18 | Evolution over time for anti-CS antibodies (full length) per protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | Specific |
| Template 16 | Comparison of the log-transformed means of the anti-CS (full length) antibodies at post-vaccination and at the time of the challenge of each vaccination schedule versus AduFx | Post-text | specific |

| Template # | Table / Figure Title | Output | Template name |
|---|---|---|---|
| | groups (Per protocol set for analysis of immunogenicity and efficacy) | destination | |
| Template 16 | Comparison of the log-transformed means of the anti-CS antibodies (full length) at post-vaccination and at the time of the challenge between Protected and Non-Protected groups (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | specific |
| Anti-CS antibo | | 1 | |
| Template 14 | Number and percentage of subjects with anti-CS (C-term) equal or above 100 EPT and GMTs (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | TIS1GMT |
| Template 14 | Number and percentage of subjects with anti-CS (C-term) equal or above 100 EPT and GMTs by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | TIS1GMT |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (C-term) at post-vaccination (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (C-term) at post-vaccination by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (C-term) at the time of the challenge (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-CS antibodies (C-term) at the time of the challenge by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 17 | Box and whiskers plot of anti-CS antibodies (C-term) at post-vaccination and the day of the challenge (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | Specific |
| Template 17 | Box and whiskers plot of anti-CS antibodies (C-term) at post-vaccination and the day of the challenge by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | Specific |
| Template 18 | Evolution over time for anti-CS antibodies (C-term) by group (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | Specific |
| Template 18 | Evolution over time for anti-CS antibodies (C-term) per protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | Specific |
| Template 16 | Comparison of the log-transformed means of the anti-CS (C-term) antibodies at post-vaccination and at the time of the challenge of each vaccination schedule versus AduFx groups (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | specific |
| Template 16 | Comparison of the log-transformed means of the anti-CS antibodies (C-term) at post-vaccination and at the time of the challenge between Protected and Non-Protected groups (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | specific |

| Template # | Table / Figure Title | Output | Template name |
|---|---|---|---|
| | | destination | |
| Anti-CS Avidity | Index (repeat) | | |
| Template 16 | Comparison of the log-transformed means of the anti-CS | Post-text | Specific |
| | avidity index (repeat) at post-vaccination and at the time of | | |
| | the challenge of each vaccination schedule versus AduFx | | |
| | groups (Per protocol set for analysis of immunogenicity and | | |
| Template 16 | efficacy) Comparison of the log-transformed means for anti-CS | Post-text | Specific |
| remplate 10 | avidity index (repeat) at post-vaccination and at the time of | FUSI-lext | Specific |
| | the challenge on Protected and Non-Protected groups (Per | | |
| | protocol set for analysis of immunogenicity and efficacy) | | |
| Template 17 | Box and whiskers plot of anti-CS avidity index (repeat) at | Post-text | Specific |
| | post-vaccination and at the time of the challenge (Per | | ' |
| | protocol set for analysis of immunogenicity and efficacy) | | |
| Template 17 | Box and whiskers plot of anti-CS avidity index (repeat) at | Post-text | Specific |
| | post-vaccination and at the time of the challenge per | | |
| | protection status (Per protocol set for analysis of | | |
| | immunogenicity and efficacy) | | |
| Anti-CS Avidity | Index post dose (full length) | | |
| Template 16 | Comparison of the log-transformed means of the anti-CS | Post-text | Specific |
| remplate to | avidity index (full length) at post-vaccination and at the time | 1 OOL LOX | Орсото |
| | of the challenge of each vaccination schedule versus AduFx | | |
| | groups (Per protocol set for analysis of immunogenicity and | | |
| | efficacy) | | |
| Template 16 | Comparison of the log-transformed means for anti-CS | Post-text | Specific |
| | avidity index (full length) at post-vaccination and at the time | | |
| | of the challenge on Protected and Non-Protected groups | | |
| | (Per protocol set for analysis of immunogenicity and | | |
| Template 17 | efficacy) Box and whiskers plot of anti-CS avidity index (full length) at | Post-text | Specific |
| remplate 17 | post-vaccination and at the time of the challenge (Per | Post-lext | Specific |
| | protocol set for analysis of immunogenicity and efficacy) | | |
| Template 17 | Box and whiskers plot of anti-CS avidity index (full length) at | Post-text | Specific |
| rompiato 17 | post-vaccination and at the time of the challenge per | 1 oot toxt | Оробіно |
| | protection status (Per protocol set for analysis of | | |
| | immunogenicity and efficacy) | | |
| | Index post dose (C-term) | _ | |
| Template 16 | Comparison of the log-transformed means of the anti-CS | Post-text | Specific |
| | avidity index (C-term) at post-vaccination and at the time of | | |
| | the challenge of each vaccination schedule versus AduFx | | |
| | groups (Per protocol set for analysis of immunogenicity and | | |
| Template 16 | efficacy) Comparison of the log-transformed means for anti-CS | Post-text | Specific |
| remplate 10 | avidity index (C-term) at post-vaccination and at the time of | FUSI-IUXI | Specific |
| | the challenge on Protected and Non-Protected groups (Per | | |
| | protocol set for analysis of immunogenicity and efficacy) | | |
| Template 17 | Box and whiskers plot of anti-CS avidity index (C-term) at | Post-text | Specific |
| p | post-vaccination and at the time of the challenge (Per | | |
| | protocol set for analysis of immunogenicity and efficacy) | | |
| Template 17 | Box and whiskers plot of anti-CS avidity index (C-term) at | Post-text | Specific |
| | post-vaccination and at the time of the challenge per | | |
| | protection status (Per protocol set for analysis of | | |
| | immunogenicity and efficacy) | | |

# 205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

| Template # | Table / Figure Title | Output destination | Template name |
|---|---|---|---|
| Anti-HBs antib | Anti-HBs antibodies | | |
| Template 14 | Number and percentage of subjects with anti-HBs equal or above 6.2 and 10 mlU/ml and GMCs (Per protocol set for analysis of immunogenicity and efficacy) | Post-text / in-<br>text / Web<br>disclosure | TIS1GMT |
| Template 14 | Number and percentage of subjects with anti-HBs equal or above 6.2 and 10 mlU/ml and GMCs by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | TIS1GMT |
| Template 15 | Reverse cumulative distribution curve for anti-HBs antibodies at post-vaccination (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-HBs antibodies at the time of the challenge (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-HBs antibodies at post-vaccination by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |
| Template 15 | Reverse cumulative distribution curve for anti-HBs antibodies at the time of the challenge by protection status (Per protocol set for analysis of immunogenicity and efficacy) | Post-text | FIS1REVCUM |

# 12.4. Reactogenicity and Safety

| Template # | Table / Listing Title | Output destination | Template name |
|---|---|---|---|
| Template 19 | Compliance in completing solicited adverse events information (Intent-to-treat set) | Post-text | TEX1COMPLIA<br>NCE |
| Template 20 | Summary of adverse events (solicited and unsolicited) within 7 days following each vaccination and overall (Intent to treat set) | In-text / Post-<br>text/Synopsis | TAC1LOCGEN |
| Template 20 | Summary of grade 3 adverse events (solicited and unsolicited) within 7 days following each vaccination and overall (Intent to treat set) | Post-text | TAC1LOCGEN |
| Template 20 | Summary of adverse events (solicited and unsolicited) with causal relationship to vaccination within 7 days following each vaccination and overall (Intent to treat set) | Post-text | TAC1LOCGEN |
| Template 20 | Summary of grade 3 adverse events (solicited and unsolicited) with causal relationship to vaccination within 7 days following each vaccination and overall (Intent to treat set) | Post-text | TAC1LOCGEN |
| Template 20 | Summary of adverse events (solicited and unsolicited) within 30 days following each vaccination and overall (Intent to treat set) | Post-text | TAC1LOCGEN |
| Template 20 | Summary of grade 3 adverse events (solicited and unsolicited) within 30 days following each vaccination and overall (Intent to treat set) | Post-text | TAC1LOCGEN |
| Template 20 | Summary of adverse events (solicited and unsolicited) with causal relationship to vaccination within 30 days following each vaccination and overall (Intent to treat set) | Post-text | TAC1LOCGEN |
| Template 20 | Summary of grade 3 adverse events (solicited and unsolicited) with causal relationship to vaccination within 30 days following each vaccination and overall (Intent to treat set) | Post-text | TAC1LOCGEN |

| Template # | Table / Listing Title | Output | Template |
|---|---|---|---|
| | | destination | name |
| Template 21 | Percentage of subject with solicited local symptoms within 7 | Post-text / | TCEMAX1FRE |
| | days following each vaccination and overall (Intent to treat | Web | QSEV |
| <del>-</del> | set) | disclosure | 051411/45450 |
| Template 31 | Bar graph of the daily prevalence of pain between day 1 and | Post-text | CEMAX1BARG |
| | day 7 following each vaccination (Intent to treat set) | | RAPH |
| Template 31 | Bar graph of the daily prevalence of redness between day 1 | Post-text | CEMAX1BARG |
| | and day 7 following each vaccination (Intent to treat set) | | RAPH |
| Template 31 | Bar graph of the daily prevalence of swelling between day 1 | Post-text | CEMAX1BARG |
| | and day 7 following each vaccination (Intent to treat set) | | RAPH |
| Template 21 | Percentage of subject with solicited general symptoms | Post-text / | TCEMAX1FRE |
| | within 7 days following each vaccination and overall (Intent | Web | QSEV |
| | to treat set) | disclosure | |
| Template 31 | Bar graph of the daily prevalence of fatigue between day 1 | Post-text | CEMAX1BARG |
| • | and day 7 following each vaccination (Intent to treat set) | | RAPH |
| Template 31 | Bar graph of the daily prevalence of gastrointestinal | Post-text | CEMAX1BARG |
| | between day 1 and day 7 following each vaccination (Intent | | RAPH |
| | to treat set) | | |
| Template 31 | Bar graph of the daily prevalence of headache between day | Post-text | CEMAX1BARG |
| rompiato o r | 1 and day 7 following each vaccination (Intent to treat set) | 1 oot toxt | RAPH |
| Template 22 | Percentage of subjects with temperature by maximum | Post-text | TCEMAX1TEM |
| Tomplate 22 | value, within 7 days following each vaccination and overall | 1 oot toxt | P |
| | (Intent to treat set) | | ' |
| Template 31 | Bar graph of the daily prevalence of temperature between | Post-text | CEMAX1BARG |
| remplate or | day 1 and day 7 following each vaccination (Intent to treat | 1 OSI-IGAL | RAPH |
| | set) | | IVALII |
| Template 30 | Summary of subjects taking a concomitant medication within | Post-text | specific |
| remplate 30 | | POSI-lext | specific |
| | 7-day following each vaccination and overall (Intent to treat | | |
| Tamplete 20 | Set) | Doot toyt | onosifio |
| Template 30 | Summary of subjects taking a concomitant medication | Post-text | specific |
| Tamanlata 02 | during the challenge phase (Intent to treat set) Summary of subjects with at least one unsolicited adverse | Doot tout / | TATACOCOT |
| Template 23 | | Post-text / | TAE1SOCPT |
| | event classified by MedDRA Primary System Organ Class | Web | |
| | and Preferred Term within 30 days of any vaccination | disclosure | |
| T I. ( . OF | (Intention-to-treat set) | D. II. I | TAE4000DT0 |
| Template 25 | Summary of subjects with unsolicited adverse events within | Post-text | TAE1SOCPTS |
| | 30 days of any vaccination by category (Intention-to-treat | | UMMARY |
| T 1 1 00 | set) | D ( ) | TAE4000DT |
| Template 23 | Summary of subjects with at least one grade 3 unsolicited | Post-text | TAE1SOCPT |
| | adverse evens classified by MedDRA Primary System | | |
| | Organ Class and Preferred Term within 30 days of any | | |
| | vaccination (Intention-to-treat set) | | |
| Template 23 | Summary of subjects with at least one related unsolicited | Post-text | TAE1SOCPT |
| | adverse event classified by MedDRA Primary System Organ | | |
| | Class and Preferred Term within 30 days of any vaccination | | |
| | (Intention-to-treat set) | | |
| Template 23 | Summary of subjects with at least one grade 3 related | Post-text | TAE1SOCPT |
| | unsolicited adverse event classified by MedDRA Primary | | |
| | System Organ Class and Preferred Term within 30 days of | | |
| | any vaccination (Intention-to-treat set) | | |
| Template 23 | Summary of subjects with at least one unsolicited adverse | Post-text/ Web | TAE1SOCPT |
| | event classified by MedDRA Primary System Organ Class | disclosure | |
| | | | i . |
| | and Preferred Term within 30 days post- challenge (Intention-to-treat set) | | |

| Template # | Table / Listing Title | Output destination | Template name |
|---|---|---|---|
| Template 23 | Summary of subjects with at least one grade 3 unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term within 30 days post- challenge (Intention-to-treat set) | Post-text | TAE1SOCPT |
| Template 23 | Summary of subjects with at least one related unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term within 30 days post- challenge (Intention-to-treat set) | Post-text | TAE1SOCPT |
| Template 23 | Summary of subjects with at least one grade3 related unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term within 30 days post- challenge (Intention-to-treat set) | Post-text | TAE1SOCPT |
| Template 25 | Summary of subjects with unsolicited adverse events within the 30 days post-challenge by category (Intention-to-treat set) | Post-text | TAE1SOCPTS<br>UMMARY |
| Template 26 | Listing of potential immune mediated disorders (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment (Intention-to-treat set) | Post-text /<br>Web<br>disclosure | TAE1PIMDLIS<br>T |
| Template 26 | Listing of meningitis reported as identified by predefined list of preferred terms and/or by investigator assessment (Intention-to-treat set) | Post-text /<br>Web<br>disclosure | TAE1PIMDLIS<br>T |

| Template # | Table / Listing Title | Output destination | Template name |
|---|---|---|---|
| Template 23 | Summary of subjects with at least one serious unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term within 30 days of any vaccination (Intention-to-treat set) | Post-text/ Web disclosure | TAE1SOCPT |
| Template 23 | Summary of subjects with at least one serious fatal unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term within 30 days of any vaccination (Intention-to-treat set) | Post-text/ Web disclosure | TAE1SOCPT |
| Template 23 | Summary of subjects with at least one serious related unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term within 30 days of any vaccination (Intention-to-treat set) | Post-text/ Web disclosure | TAE1SOCPT |
| Template 23 | Summary of subjects with at least one serious unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term occurring from Dose 1 (Day 1) until the last study visit (Day 376) (Intention-to-treat set) | Post-text /<br>Web<br>disclosure | TAE1SOCPT |
| Template 24 | Summary of occurrences and subjects with at least one serious unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term occurring from Dose 1 (Day 1) until the last study visit (Day 376) (Intention-to-treat set) | Web<br>disclosure | TAC1SOCPT |
| Template 23 | Summary of subjects with at least one serious fatal unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term occurring from Dose 1 (Day 1) until the last study visit (Day 376) (Intention-to-treat set) | Post-text /<br>Web<br>disclosure | TAE1SOCPT |
| Template 23 | Summary of subjects with at least one serious related unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term occurring from Dose 1 (Day 1) until the last study visit (Day 376) (Intention-to-treat set) | Post-text/ Web disclosure | TAE1SOCPT |
| Template 23 | Summary of subjects with at least one serious unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term occurring from day of challenge until the end of challenge phase (Day 314) (Intention-to-treat set) | Post-text /<br>Web<br>disclosure | TAE1SOCPT |
| Template 23 | Summary of subjects with at least one serious fatal unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term occurring from day of challenge until the end of challenge phase (Day 314) (Intention-to-treat set) | Post-text/ Web disclosure | TAE1SOCPT |
| Template 23 | Summary of subjects with at least one serious related unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term occurring from day of challenge until the end of challenge phase (Day 314) (Intention-to-treat set) | Post-text/ Web disclosure | TAE1SOCPT |
| Template 27 | Listing of SAEs reported from study start to end of the study (Intention-to-treat population) | Post-text | TAE1SAELIST |
| Template 28 | Listing of (S) AEs and solicited symptoms leading to study/treatment discontinuation (Intent to treat set) | Post-text /<br>Web<br>disclosure/ | TAE1WITHDR<br>AWAL |

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

| Template # | Table / Listing Title | Output destination | Template name |
|---|---|---|---|
| Template 24 | Summary of occurrences and subjects with at least one solicited or unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term (excluding the SAEs) occurring within 30 days of any vaccination (Intention-to-treat set) | Web<br>disclosure | TAC1SOCPT |
| Template 29 | Summary of hematology and biochemistry results (Intention-to-treat population) | Post-text/ Web disclosure | TLB1RANGEV<br>SBSL |

# 12.5. Individual data listings:

Reason for non-eligibility (LIE1LIST)

Demography (LDM1DEMOG)

Reason for visit not done (LDS1NOVIS)

Immunogenicity (LIS1LIST)

Vaccine administration (LEC1EXPO)

Reason for vaccine not administered (LEC1NOADM)

Solicited local adverse events (LEC1LOC)

Solicited general adverse events (LEC1GEN)

Concomitant medications (LCM1LIST)

Pregnancy (Specific)

# 12.6. Template of tables, figures AND LISTINGS

# 12.6.1. Demographics and baseline characteristics

## Template 1 Consort flow (Enrolled set)

| | | otal<br>=xx |
|--------------------------------------------------|---|-------------|
| | n | % |
| NUMBER OF SUBJECTS WHO SIGNED INFORMED CONSENT | | |
| NUMBER OF SUBJECTS WITHDRAWN PRIOR TO | | |
| RANDOMIZATION | | |
| Consent Withdrawal, Not Due To A Serious Adverse | | |
| Event and/or An Adverse Event | | |
| Eligibility Criteria Not Fulfilled | | |
| Lost To Follow-Up | | |
| Migrated / Moved From The Study Area | | |
| Missing | | |
| Other | | |
| NUMBER OF SUBJECTS INCLUDED IN RANDOMIZED | | |
| SET (=INTENT-TO-TREAT SET) | | |
| | | · |

N = Number of subjects who have signed ICF (screened)

Withdrawal reason "Other" corresponds to Subject Enrollment target reached before Randomization

**Template 2** Consort flow (Intent to treat set)

| | <gro<br>N=)<br/>N</gro<br> | up 1><br>(XX<br>% | <group<br>N=XX<br/>N 9</group<br> | | Total<br>N=XXX<br>N | <b>(</b><br>% |
|---|---|---|---|---|---|---|
| Number of subjects eliminated from per protocol set | xxx | 100 | xxx | 100 | xxx | 100 |
| <elimination 1<br="" reason="">(code)&gt;<br/><elimination 2<="" reason="" td=""><td></td><td></td><td></td><td></td><td></td><td></td></elimination></elimination> | | | | | | |
| (code)> | XXXX | | XXXX | | XXXX | |
| | XXX | | XXX | | xxxx | |
| Number of subjects included in PPS | XXXX | X.XX | XXX | X.XX | XXX | X.XX |

Short group label = long group label

N = total number of subjects randomized

n/% = number / percentage of subjects in a given category

<sup>% =</sup> n / Number of subjects with available results x 100

All Enrolled Set includes Screen Failures and non-Randomized subjects.

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

Summary of visit attendance (Intent-to treat set) Template 3

| | | <group 1=""><br/>N=XXXX</group> | | <group xxx=""><br/>N=XXXX</group> | | tal<br>XXXX |
|---|---|---|---|---|---|---|
| | n | % | n | % | n | % |
| Visit 1 (Day 1) | | | | | | |
| Attended | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Did not attend yet | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Withdrawal at visit or earlier | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Did not attend | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Visit 2 (Day xx) | | | | | | |
| Visit 3 (Day xx) | | | | | | |
| Last study contact (Day 376) | | | | | | |
| Completed | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Did not complete yet | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Withdrawal at visit or earlier | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Did not complete | XXX | XX.X | XXX | XX.X | XXX | XX.X |

Template 4 Summary of disposition <analysis set name>

| | | <group 1=""><br/>N=XXXX</group> | | <group 2=""><br/>N=XXXX</group> | | otal<br>XXXX |
|---|---|---|---|---|---|---|
| | n | % | n | % | n | % |
| Completed the study | xxx | XX.X | XXX | XX.X | XXX | XX.X |
| Primary reason for withdrawal | | | | | | |
| DEATH | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| ADVERSE EVENT | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| PROTOCOL DEVIATION | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| WITHDRAWAL BY SUBJECT | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| MIGRATED / MOVED FROM THE STUDY AREA | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| LOST TO FOLLOW-UP | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| STUDY TERMINATED BY SPONSOR | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| OTHER | XXX | XX.X | XXX | XX.X | XXX | XX.X |

Short group label = long group label

N = total number of subjects

n/% = number / percentage of subjects in a given category
Note: the list of reasons will be study specific

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

Template 5 Summary of important protocol deviations leading to elimination <analysis set name>

| Category | <group 1=""></group> | | <gr< th=""><th colspan="2"><group 2=""></group></th><th colspan="3">Total</th></gr<> | <group 2=""></group> | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|
| Sub-category | осс | n | % | осс | n | % | осс | n | % |
| At least one important protocol deviation | xxx | XXX | XX.X | xxx | XXX | xx.x | xxx | xxx | XX.X |
| <category 1=""></category> | XXX | XXX | XX.X | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <sub-category 1=""></sub-category> | XXX | XXX | XX.X | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <sub-category 2=""></sub-category> | XXX | XXX | XX.X | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <category 2=""></category> | XXX | XXX | XX.X | XXX | xxx | XX.X | XXX | XXX | XX.X |

Short group label = long group label
Occ = number of occurrences = number of important protocol deviations

n/% = number / percentage of subjects in a given category

Note: Categories presented by occurrence frequency and within categories the sub-categories will be sorted by occurrence frequency. For a same frequency then sorted alphabetically

 05-DEC-2018

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

Template 6 Deviations from protocol for age and intervals between study visits <analysis set name>

| Type of interval | Interval range | <group 1=""></group> | | | <group th="" x<=""><th>xx&gt;</th></group> | xx> | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Value | % | V | alue | % |
| Age (years) at first vaccine | From <x> to <y> years</y></x> | N | | XXX | | XXX | | |
| administration | | n | | XXX | | XXX | XX.X | |
| | | Below <x></x> | XX.X | | | XXX | XX.X | |
| | | Above <y></y> | | XXX | | XXX | XX.X | |
| | | · | XX.X | | | | | |
| Number of days between | From <x> to <y> days</y></x> | | | XXX | | | | |
| vaccination <x> and vaccination <y></y></x> | | | XX.X | | | | | |
| Number of days between vaccination <x> and visit <y></y></x> | From <x> to <y> days</y></x> | | | | | | | |
| • | From <x> to <y> days</y></x> | | | | | | | |
| Number of days between vaccination <x> and blood sampling <y></y></x> | , , | | | | | | | |

05-DEC-2018 

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

Template 7 Summary of demographic characteristics <analysis set name>

| | <each group=""></each> | |
|---|---|---|
| | Value or n | N=XXXX<br>% |
| Age (years) at first vaccination/screening (for cor | | 7 |
| n | , XXX | |
| Mean | XXX.X | |
| Standard Deviation | XXX.X | |
| Median | XXX.X | |
| Minimum | XXX | |
| Maximum | XXX | |
| Sex | | |
| Male | XXX | XX.X |
| Female | XXX | XX.X |
| Race | | |
| American indian or alaska native | XXX | XX.X |
| Asian | XXX | XX.X |
| Black or african american | XXX | XX.X |
| Native hawaiian or other pacific islander | XXX | XX.X |
| White | XXX | XX.X |
| Other | XXX | XX.X |

Short group label = long group label n/% = number / percentage of subjects in a given category

 05-DEC-2018

Template 8 Summary of demography and baseline characteristics <Enrolled Set>

| | Total<br>N=XXXX | |
|---|---|---|
| | Value or n | <b>`</b> |
| Age ( <days months="" weeks="" years="">) at first vaccination</days> | | |
| n | XXX | |
| Mean | XXX.X | |
| Standard Deviation | XXX.X | |
| Median | XXX.X | |
| Minimum | XXX | |
| Maximum | XXX | |
| Age group [EudraCT] | | |
| Adults (18-64 years) | XXX | XX.X |
| Country<br>USA | xxx | XX.X |
| <br>Sex | | |
| Male | XXX | XX.X |
| Female | XXX | XX.X |
| Race | | |
| American Indian Or Alaska Native | XXX | XX.X |
| Asian | XXX | XX.X<br>XX.X |
| Black Or African American | XXX | XX.X |
| Native Hawaiian Or Other Pacific Islander | XXX | XX.X |
| White | XXX | XX.X |
| Other | XXX | XX.X |

05-DEC-2018 

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

# Template 9 Summary of previous Hepatitis B vaccination (Intent-to-treat set)

| | | <each group=""></each> |
|---|---|---|
| | | N=XXXX |
| , | Value or n | % |
| Subjects with an history of Hepatitis B vaccination | XXXXX | XXXX |
| Subjects without an history of Hepatitis B vaccination | XXX | XXXXX |

Short group label = long group label

n/% = number / percentage of subjects in a given category

## Template 10 Exposure to study vaccine by visit (Intent-to-treat)

| | Vaccine administered | <group 1=""><br/>N=XXX</group> | <group 2=""><br/>N=XXX</group> |
|---|---|---|---|
| | | n % | n % |
| Visit 2 (Day 1) | <vaccine 1=""></vaccine> | XXX XX.X | XXX XX.X |
| | <vaccine 2=""></vaccine> | xxx xx.x | XXX XX.X |
| Visit 3 (Day 28) | | | |

. . .

Short group label = long group label

n/% = number / percentage of subjects in a given category

05-DEC-2018 

# **12.6.2.** Efficacy

Template 11 Parasitemia incidence defined by a positive blood slide and vaccine efficacy versus control of <each group> (Per protocol set for analysis of immunogenicity and efficacy)

| | <group 1=""></group> | <group xxx=""></group> |
|------------|----------------------|------------------------|
| | N=XXXX | N=XXXX |
| arasitemia | n xx.x | xx.x |
| | % xxxx | XXXX |
| | 95% CI (xx.x; xx.x) | (xx.x; xx.x) |
| | p-value xx.x | XX.X |
| | (versus xxx) | |

Short group label = long group label

N = number of subjects included in each group (without missing values)

n/% = number / percentage of subjects reporting at least one event(s) in each group

LL, UL = 95% Lower and Upper confidence limits

P-value from Fisher's Exact test (computed versus control or AduFx group)

05-DEC-2018 

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

Template 12 Time to onset of parasitemia by blood slide (Per protocol set for analysis of immunogenicity and efficacy)

| | | <each group=""></each> |
|----------------------|--------|------------------------|
| | N=XXXX | |
| | Value | |
| | or n | % |
| Time to onset (days) | | |
| n | XXX | |
| Mean | XXX.X | |
| Standard Deviation | XXX.X | |
| Median | XXX.X | |
| Minimum | XXX | |
| Maximum | XXX | |
| p-value (versus xx) | XXXX | |

Short group label = long group label

Template 13 Cumulative incidence of parasitemia onset defined by positive blood slide for all groups (Per protocol set for analysis of immunogenicity and efficacy)

Figure 1 Kaplan-Meier curve for time to onset of parasitemia following primary challenge: RTS,S/AS02A vs RTS,S/AS01B - pooled Cohorts 1 and 2



----- = RTS,S/AS02A; ----- = RTS,S/AS01B; o = censored

05-DEC-2018 

# 12.6.3. Immunogenicity

Template 14 Number and percentage of subjects with <assay description> equal or above <cut-off> and GMCs (Per protocol set for analysis of immunogenicity and efficacy)

| Antibody | Time point | Cut-off | | | | <0 | roup 1 | > | | | <group 2=""></group> | | | | | <group 3=""></group> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | 95% CI | | | 95% CI | | | | | | 95 | % CI | |
| | | | | N | n | value | LL | UL | N | n | value | LL | UL | N | n | value | LL | UL |
| <antibody 1<="" td=""><td>&gt; <time point<="" td=""><td>1&gt; <cut-off 1=""></cut-off></td><td>%&gt;=<cut-off 1=""> <unit></unit></cut-off></td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td></time></td></antibody> | > <time point<="" td=""><td>1&gt; <cut-off 1=""></cut-off></td><td>%&gt;=<cut-off 1=""> <unit></unit></cut-off></td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td></time> | 1> <cut-off 1=""></cut-off> | %>= <cut-off 1=""> <unit></unit></cut-off> | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| • | • | | %>= <cut-off 2=""> <unit></unit></cut-off> | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | | %>= <cut-off 3=""> <unit></unit></cut-off> | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | | GM <t,c></t,c> | XXX | | XX.X | XX.X | XX.X | XXX | | XX.X | XX.X | XX.X | xxx | | XX.X | XX.X | XX.X |

GMC = geometric mean concentration

N = number of subjects with available results

n/% = number/percentage of subjects with concentration within the specified range

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit;

05-DEC-2018 

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

Template 15 Reverse cumulative distribution curve for <assay description> <timing> (Per protocol set for analysis of immunogenicity and efficacy)

#### Example:



Short group label = long group label

#### All groups at one timepoint

Template 16 Comparison of the log-transformed means of the <anti-CS> antibodies <repeat/full-length/C-term> at post-vaccination of <each vaccination schedule versus AduFx / Protected versus Non-protected> (Per protocol set for analysis of immunogenicity and efficacy)

| | | <each group=""></each> |
|---------------------|-------|------------------------|
| | | N=XXXX |
| | Value | |
| | or n | % |
| < timing > | | |
| N | XXX | |
| Mean | XXX.X | |
| 95% of the mean | | |
| Standard Deviation | XXX.X | |
| Median | | |
| Q1 | | |
| Q3 | | |
| Minimum | | |
| Maximum | | |
| p-value (versus xx) | | |
| < timing > | | |

N = number of subjects with available results

Note: for Mean, also display the 95% CI

Timing: post-dose 2 or 2 and day of challenge (in the same table)

Template 17 Box and whiskers plot of <assay description> <timing> (Per protocol set for analysis of immunogenicity and efficacy)

# Example:



Template 18 Evolution over time for <assay descrition (Per protocol set for analysis of immunogenicity and efficacy)



205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

#### Reactogenicity and safety 12.6.4.

Template 19 Compliance in completing solicited adverse events information (intent-to-treat)

| | | | <group 1=""></group> | • | Group 2> | |
|---|---|---|---|---|---|---|
| | | N | n | N | n | Compliance |
| | | Compli | ance | | | (%) |
| | | (%) | | | | |
| <vaccination at<="" td=""><td>General solicited adverse</td><td>XXX</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td></vaccination> | General solicited adverse | XXX | XX.X | XXX | XXX | XX.X |
| visit 1> | events | XXX | XX.X | XXX | XXX | XX.X |
| | Local solicited adverse | XXX | | | | |
| | events | XXX | XX.X | XXX | XXX | XX.X |
| <vaccination at<="" td=""><td></td><td></td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td></vaccination> | | | XX.X | XXX | XXX | XX.X |
| visit X> | General solicited adverse | XXX | | | | |
| | events | XXX | | | | |
| | Local solicited adverse | XXX | | | | |
| | events | XXX | XX.X | XXX | XXX | XX.X |
| | | | XX.X | XXX | XXX | XX.X |
| Per vaccination | | | | | | |
| | General solicited adverse | XXX | | | | |
| | events | XXX | | | | |
| | Local solicited adverse | XXX | | | | |
| | events | XXX | | | | |

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

Template 20 Incidence and nature of symptoms (solicited and unsolicited) within 7-day following each vaccination and overall (Intention-to-treat set)

| | | | <gro< th=""><th>up 1&gt;</th><th></th><th></th><th><grot< th=""><th colspan="4"><group 2=""></group></th></grot<></th></gro<> | up 1> | | | <grot< th=""><th colspan="4"><group 2=""></group></th></grot<> | <group 2=""></group> | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | 95 | % CI | | | 95% CI | |
| | | n | % | LL | UL | n | % | LL | UL |
| <vaccination 1="" at="" visit=""> N</vaccination> | | XXX | | | | XXX | | | |
| | Any symptom | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Local symptom | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | General symptom | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |

<Vaccination at visit 2> ...

. . .

Per subject

Per vaccination

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects presenting at least one type of symptom whatever the study vaccine administered

For overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom whatever the study vaccine administered 95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

Template 21 Incidence of solicited <local/general> symptoms within 7-day following each vaccination and overall (Intention-to-treat set)

Symptom: Xxxxx

| | | | <gro< th=""><th>up 1&gt;</th><th></th><th></th><th><grot< th=""><th colspan="2">ıp 2&gt;</th></grot<></th></gro<> | up 1> | | | <grot< th=""><th colspan="2">ıp 2&gt;</th></grot<> | ıp 2> | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% CI | | | | | |
| | | n | % | LL | UL | n | % | LL | UL |
| <vaccination 1="" at="" visit=""></vaccination> | N | XXX | | | | XXX | | | |
| | Any | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Related | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Grade 3 | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Grade 3 related | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Medically attended visit | | | | | | | | |

<Vaccination at visit 2> ...

Per subject

#### Per vaccination

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects reporting at least once the symptom

For Overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom

Total : n/%= number/percentage of subjects/doses with at least one local symptom whatever the number of injections.

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

Template 22 Incidence of temperature by maximum value, within 7 days following each vaccination and overall (Intention-to-treat set)

| | _ | | <gro< th=""><th>up 1&gt;</th><th></th><th>•</th><th><gro< th=""><th>ıp 2&gt;</th><th><u> </u></th></gro<></th></gro<> | up 1> | | • | <gro< th=""><th>ıp 2&gt;</th><th><u> </u></th></gro<> | ıp 2> | <u> </u> |
|---|---|---|---|---|---|---|---|---|---|
| | | | | 95 | % CI | | | 959 | <b>6 CI</b> |
| | | n | % | LL | UL | n | % | LL | UL |
| <vaccination 1="" at="" visit=""></vaccination> | N<br>≥37.5 | XXX | | | | XXX | | | |
| | <39.0 | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | related | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | <39.0 related | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| <vaccination 2="" at="" visit=""></vaccination> | | | | | | | | | |
| Per subject | | | | | | | | | |
| Per vaccination | | | | | | | | | |

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

Template 23 Summary of <subjects with/ vaccinations followed by> at least one <serious/related/related serious/fatal> unsolicited adverse events <medically attended visits>, <within 30 days of any vaccination/ within 30 days of post-challenge period / from study start to 30 days post-challenge> (Intention-to-treat set)

| | | <gro< th=""><th>up 1&gt;</th><th></th><th></th><th colspan="5"><group 2=""></group></th></gro<> | up 1> | | | <group 2=""></group> | | |
|---|---|---|---|---|---|---|---|---|
| | | N=X | XXX | | | N=X | XXX | |
| Primary System Organ Class (CODE) | | | 95 | % CI | | | 959 | % CI |
| Preferred Term (CODE) | n | % | LL | UL | n | % | LL | UL |
| Any <Ø, serious, related, related serious, fatal> unsolicited adverse event <Ø, - Medically Attended Visits> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| <soc (code)="" 1=""></soc> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| <preferred (code)="" 1="" term=""></preferred> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| <preferred (code)="" 2="" term=""></preferred> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| <soc (code)="" 2=""></soc> | xxx | XX.X | xx.x | XX.X | XXX | XX.X | XX.X | XX.X |
| <preferred (code)="" 1="" term=""></preferred> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| <preferred (code)="" 2="" term=""></preferred> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |

At least one symptom = At least one symptom experienced regardless of the System Organ Class

95% CI = Exact 95% confidence interval

Template 24 Summary of occurrences and subjects with at least one serious unsolicited adverse events from study start until last study visit (D314) (Intention-to-treat set)

| Primary System Organ Class (CODE) | | Group 1<br>N=XXXX | | <group xxx=""><br/>N=XXXX</group> | | |
|---|---|---|---|---|---|---|
| Preferred Term (CODE) | осс | n | % | осс | n | % |
| Any < $\emptyset$ , serious, related serious, fatal, related fatal> < $\emptyset$ , solicited and> unsolicited adverse event | XXX | XXX | XX.X | XXX | xxx | XX.X |
| <soc (code)="" 1=""></soc> | XXX | xxx | XX.X | XXX | XXX | XX.X |
| <preferred (code)="" 1="" term=""></preferred> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <preferred (code)="" 2="" term=""></preferred> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <soc (code)="" 2=""></soc> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <preferred (code)="" 1="" term=""></preferred> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <preferred (code)="" 2="" term=""></preferred> | XXX | XXX | XX.X | XXX | XXX | XX.X |

N = Number of subjects having received at least one dose

n/% = Number / percentage of subjects reporting at least once a specified symptom within 30 days after vaccination day 0 to day 29

205081 (MALARIA-092) Statistical Analysis Plan Amendment 1 Final

Template 25 Summary of subjects by unsolicited event category, <within 30 days of any vaccination/ within 30 days of post-challenge period / from study start to 30 days post-challenge> (Intention-to-treat set)

| | | | up 1><br>XXX | | <group 2=""><br/>N=XXXX</group> | | | |
|---|---|---|---|---|---|---|---|---|
| | 95% CI | | | | | | 95% CI | |
| | n | % | LL | UL | n | % | LL | UL |
| At least one unsolicited adverse event | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| At least one serious unsolicited adverse event | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| At least one related unsolicited adverse event | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| At least one serious related unsolicited adverse event | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |

Template 26 Listing of potential immune-mediated disorders (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment (Intent to treat set)

| Group | Subject<br>number | Gender | | Country | Race | | Verbatim<br>Preferred | Verbatim<br>Preferred Term | | Primary S<br>Organ Cla | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXX | XXXXX | | XXXXXXX | xxxxxx | XX | XXXXX | | XXX | | | XXXXX |
| Group | • | | Medical | Vaccination | • | | Duration | Intensity | | Outcome | | pIMD |
| | number | | visit type | | onset | | | Causality | | | (Y/N) | Source |
| XXXXX | xxxxx | | xxxxxx | XXXXXX | XX | | XX | XXXX | XXX | XXXXX | XX | xxxxx |

Template 27 Listing of SAEs reported from study start to 28 days post challenge (Intention-to-treat set)

| Group | Subject<br>number | Gender | Country | Race | Age at<br>onset<br>(Year) | Verbatim | | Preferred 1 | Term | |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXX | XXXXX | XXXXXXX | XXXXXX | XX | XXXXX | | XXXXX | | |
| Group | Subject<br>number | Primary<br>System<br>Organ<br>Class | | Medical<br>visit type | Vaccinati<br>on | Day of<br>onset | Duration | Intensity<br>Causality | | Outcome |
| XXXXX | XXXXX | XXXXX | | XXXXXXX | XXXXXX | XX | XX | XXXX | XXX | XXXXX |

205081 (MALARIA-092)

Statistical Analysis Plan Amendment 1 Final

Template 28 Listing of (S) AEs and solicited symptoms leading to study/treatment discontinuation (Intent to treat set)

| | Subject<br>number | Gender | Country | | | SAE (Y/N)<br>Causality | | Vaccination and visit |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxx | xxxxx | xxxxxx | xxxxx | xxxxx | x x<br>Vaccination: | xxxx<br>x at visit x | xxxxx |

#### Template 29 Summary of hematology and biochemistry results (Intention-to-treat set)

| Timepoint | Value at timepoint | <group 1=""></group> | <group 2=""></group> |
|---|---|---|---|
| | | N % | N % |
| <timepoint 1=""></timepoint> | N | xxx | XXX |
| | Grade 1 | XXX XX.X | XXX XX.X |
| | Grade 2 | XXX XX.X | XXX XX.X |
| | Grade 3 | XXX XX.X | XXX XX.X |
| | Grade 4 | XXX XX.X | XXX XX.X |
| | Unknown | XXX XX.X | XXX XX.X |

N = Number of subjects having received at least one dose

Template 30 Summary of subjects taking a concomitant medication with <7 days following each vaccination and overall / during challenge phase> (Intent to treat set)

| | | <group 1=""></group> | | | | | <group 2=""></group> | | |
|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | | | <b>6 CI</b> | | |
| | | n | % | LL | UL | n | % | LL | UL |
| <vaccination 1="" at="" visit=""></vaccination> | N | XXX | | | | XXX | | | |
| | Any | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Any antipyretic | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |

...

Per subject

Per vaccination

n/% = Number / percentage of subjects in each category

Template 31 Bar graph of the daily prevalence of <pain/redness/swelling> between day 1 and day 7 following each vaccination (Intent to treat set)

# Example:



Template 32 Minimum and maximun dates (intent-to-treat set)

| | | <each group=""></each> | <each group=""></each> | Overall |
|---|---|---|---|---|
| Visit Description | Parameter | Date | Date | Date |
| < each informed consent> | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| [Randomization] | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| <each visit=""></each> | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |

Short group label = long group label

| | Statistical Arialysis Flatt Fillal |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A Phase IIa, open-label, controlled, mono-center study to evaluate the efficacy, immunogenicity and safety of GSK Biologicals' candidate malaria vaccines RTS,S/AS01 <sub>E</sub> and RTS,S/AS01 <sub>B</sub> administered as various dose schedules according to a 0, 1, 7-month or a 0, 7-month schedule in healthy malaria-naïve subjects aged 18-55 years. |
| eTrack study number and<br>Abbreviated Title | 205081 (MALARIA-092) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Final: 24-MAY-2018 |
| Co-ordinating author: | PPD (Statistician) |
| Reviewed by: | PPD (Clinical Research and Development Lead) PPD (Lead Scientific writer) PPD (Scientific writer) PPD (Regulatory Affair) PPD (SERM physician) PPD (SERM Scientist) PPD (CLS Manager) PPD (Lead statistical analyst) PPD (Lead statistician) PPD (Public disclosure) |
| Approved by: | PPD (Clinical Research and Development Lead) PPD (Lead Scientific writer) PPD (Lead statistical analyst) PPD (Lead statistician) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14April 2017)

205081 (MALARIA-092) Statistical Analysis Plan Final

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | T OF A | BBREVIATIONS | 6 |
| 1. | DOC | JMENT HISTORY | 8 |
| 2. | STUD | Y DESIGN | 9 |
| 2 | OD IE | CTIVES | 10 |
| 3. | 3.1. | CTIVESPrimary objective | |
| | 0.1. | 3.1.1. Efficacy | |
| | 3.2. | Secondary objectives | |
| | | 3.2.1. Efficacy | |
| | | 3.2.2. Immunogenicity | |
| | 0.0 | 3.2.3. Safety | |
| | 3.3. | Tertiary objectives | |
| | | 5.5.1. Illinunogenicity | 13 |
| 4. | ENDF | POINTS | 13 |
| | 4.1. | Primary endpoint | |
| | 4.0 | 4.1.1. Efficacy | |
| | 4.2. | Secondary endpoints | |
| | | 4.2.1. Efficacy4.2.2. Immunogenicity | |
| | | 4.2.3. Safety | |
| | 4.3. | Tertiary endpoints | |
| | | 4.3.1. Immunogenicity | |
| 5. | ΛΝΙΛΙ | YSIS SETS | 17 |
| Ο. | 5.1. | Definition | |
| | 0.1. | 5.1.1. Enrolled Set | |
| | | 5.1.2. Intent-to-treat set (ITTS) | |
| | | 5.1.3. Per-Protocol Set for analysis of immunogenicity and | |
| | | efficacy (PPS for analysis of immunogenicity and efficacy) | 17 |
| | | 5.1.4. Adapted Per-Protocol Set for analysis of efficacy (Adapted | |
| | <b>5</b> 0 | PPS for analysis of efficacy) | 17 |
| | 5.2. | Criteria for eliminating data from Analysis Sets | |
| | | 5.2.2. Elimination from the PPS for analysis of immunogenicity | 10 |
| | | and efficacy | 18 |
| | | 5.2.2.1. Excluded subjects | |
| | | 5.2.3. Elimination from the Adapted PPS for analysis of efficacy | |
| | | 5.2.3.1. Excluded subjects | 20 |
| | 5.3. | Important protocol deviations not leading to elimination from per-<br>protocol analysis set | 20 |
| | | • | |
| 6. | | ISTICAL ANALYSES | |
| | 6.1. | Demography | 21 |
| | | 6.1.1. Analysis of demographics/baseline characteristics planned | 04 |
| | 6.2. | in the protocol | |
| | 0.2. | | <u>4</u> |

## 205081 (MALARIA-092) Statistical Analysis Plan Final

| | 6.3. | 6.2.1. | Analysis of exposure planned in the protocolanalysis | 21 |
|---|---|---|---|---|
| | 0.3. | 6.3.1. | Analysis of efficacy planned in the protocol | <mark>22</mark> |
| | | 6.3.2. | Additional considerations | |
| | | | 6.3.2.1. Case definition | |
| | | | 6.3.2.2. Risk periods | |
| | 6.4. | | genicity analysis | |
| | | 6.4.1. | Analysis of immunogenicity planned in the protocol | |
| | 0.5 | 6.4.2. | Additional considerations | |
| | 6.5. | | of safety | |
| | | 6.5.1. | Analysis of safety planned in the protocol | |
| | | 6.5.2. | Additional considerations | 21 |
| 7. | ANALY | 'SIS INTE | ERPRETATION | 27 |
| 8. | COND | UCT OF A | ANALYSES | 28 |
| • | 8.1. | | e of analyses | |
| | 8.2. | | al considerations for interim analyses | |
| 9. | CHAN | GES FRO | OM PLANNED ANALYSES | 28 |
| 10. | LIST C | F FINAL | REPORT TABLES, LISTINGS AND FIGURES | 28 |
| 11. | ANNE | X 1 STAN | IDARD DATA DERIVATION RULE AND STATISTICAL | |
| | METH | ODS | | <mark>29</mark> |
| | 11.1. | | al Method References | |
| | 11.2. | | data derivationd | |
| | | 11.2.1. | | |
| | | 11.2.2. | Dose number | |
| | | 11.2.3. | Demography | |
| | | 11.2.4. | Immunogenicity | |
| | | 11.2.5. | Safety | 31 |

205081 (MALARIA-092) Statistical Analysis Plan Final

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Intervals between study visits for the investigational vaccine groups: AduFx, 2PedFx, PedFx, and Adu2Fx | 10 |
| Table 2 | Intervals between study visits for the investigational vaccine group: Adu1Fx | 10 |
| Table 3 | Intervals between study visits for the infectivity control group | 10 |
| Table 4 | Toxicity grading scales for blood testing | 26 |

205081 (MALARIA-092) Statistical Analysis Plan Final

# **LIST OF FIGURES**

| | | PAGE |
|----------|--------------|-------|
| Figure 1 | Study design | <br>9 |

205081 (MALARIA-092) Statistical Analysis Plan Final

## **LIST OF ABBREVIATIONS**

AE Adverse event

Anti-CS Antibody to the *Plasmodium falciparum* circumsporozoite (CS) repeat

domain

Anti-HBs Antibody to the hepatitis B surface antigen

AS01<sub>B</sub> GSK's proprietary Adjuvant System containing MPL, QS-21 and

liposome (50 µg MPL and 50 µg QS-21)

AS01<sub>E</sub> GSK's proprietary Adjuvant System containing MPL, QS-21 and

liposome (25 µg MPL and 25 µg QS-21)

ALT Alanine aminotransferase

AST Aspartate aminotransferase

ATP According-To-Protocol

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

CLS Clinical laboratory sciences

CRF Case Report Form

C-term CS terminal portion of the protein

CTRS Clinical Trial Registry Summary

eCRF electronic Case Report Form

EPT Endpoint titer

ES Exposed Set

EU/ml ELISA unit per milliliter

GMC Geometric mean concentration

GSK GlaxoSmithKline

HBsAg Hepatitis B surface Antigen

ICH Internal Conference on Harmonization

IgG Immunoglobulin G

IU/ml International units per milliliter

ITTS Intent-To-Treat Set

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

mIU/ml Milli International units per milliliter

NP Not protected

P Protected
205081 (MALARIA-092) Statistical Analysis Plan Final

PCR Polymerase chain reaction

PD Protocol Deviation

pIMD potential Immune Mediated Disease

PPS Per-Protocol Set

SAE Serious adverse event

SAS Statistical Analysis System

SAP Statistical Analysis Plan

SD Standard Deviation

SERM Safety Evaluation and Risk Management

SHS Study Headline Summary

TFL Tables Figures and Listings

TOC Table of Content

UL Upper Limit of the confidence interval

ULN Upper Limit of normal range

VE Vaccine Efficacy

WBC White blood cells

205081 (MALARIA-092) Statistical Analysis Plan Final

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|-------------------------------------|
| 24-MAY-2018 | Final version | Administrative Change – 19-JUN-2017 |

# 2. STUDY DESIGN

Figure 1 Study design



D: Day; Mth: month; R: RTS,S; SCR: Screening; V: visit. \* Blood sample for estimation of subjects with parasitemia (PCR testing) will be collected on the day of subject entry into the hotel phase (Day 295 [Visit 16]); blood sample for biochemistry and hematology parameters will be collected the day of first parasitemia and blood sample for assessment of parasitemia (blood smear) will be collected daily for 14 days (from Day 291 [Visit 12] to Day 304 [Visit 25]) and then every two days for nine days (Day 306 [Visit 26], Day 308 [Visit 27], Day 310 [Visit 28], Day 312 [Visit 29], and Day 314 [Visit 30]).

24-MAY-2018 Page 9 of 32

The following table gives the intervals between study visits at defined visits to apply, as described in the protocol:

Table 1 Intervals between study visits for the investigational vaccine groups: AduFx, 2PedFx, PedFx, and Adu2Fx

| Interval | Optimal length of interval <sup>1</sup> | Allowed interval <sup>2</sup> |
|---|---|---|
| Visit 1 (Screening) → Visit 2 (1st vaccination) | 0 to 90 days | - |
| Visit 2 → Visit 3 (2 <sup>nd</sup> vaccination) | 28 days | ± 7 days |
| Visit $3 \rightarrow \text{Visit } 5$ | 7 days | ± 1 day |
| Visit 3 → Visit 6 | 30 days | ± 7 days |
| Visit 3 → Visit 7 (3 <sup>rd</sup> vaccination) | 168 days | ± 14 days |
| Visit 7 → Visit 9 | 7 days | ± 1 day |
| Visit 7 → Visit 10 | 30 days | ± 7 days |
| Visit 7 → Visit 11 (Challenge) | 90 days | + 14 days |
| Visit 11 → Visit 30 | 28 days | ± 7 days |
| Visit 30 → Visit 31 | 62 days | ± 14 days |

<sup>&</sup>lt;sup>1</sup>Whenever possible the investigator should arrange study visits within this interval.

Table 2 Intervals between study visits for the investigational vaccine group: Adu1Fx

| Interval | Optimal length of interval <sup>1</sup> | Allowed interval <sup>2</sup> |
|---|---|---|
| Visit 1 (Screening) → Visit 2 (1st vaccination) | 0 to 90 days | - |
| Visit 2 → Visit 7 (2 <sup>nd</sup> vaccination) | 196 days | ± 14 days |
| Visit 7 → Visit 9 | 7 days | ± 1 day |
| Visit 7 → Visit 10 | 30 days | ± 7 days |
| Visit 7 → Visit 11 (Challenge) | 90 days | + 14 days |
| Visit 11 → Visit 30 | 28 days | $\pm$ 7 days |
| Visit 30 → Visit 31 | 62 days | $\pm$ 14 days |

<sup>&</sup>lt;sup>1</sup> Whenever possible the investigator should arrange study visits within this interval.

Table 3 Intervals between study visits for the infectivity control group

| Interval | Optimal length of interval <sup>1</sup> | Allowed interval <sup>2</sup> |
|---|---|---|
| Visit 1b (Screening) → Visit 11 (Challenge) | 0 to 56 days | - |
| Visit 11 → Visit 30 | 28 days | ± 7 days |

<sup>&</sup>lt;sup>1</sup>Whenever possible the investigator should arrange study visits within this interval.

<sup>&</sup>lt;sup>2</sup> Subjects may not be eligible for inclusion in the according-to-protocol (ATP) cohort for analysis of immunogenicity and efficacy if they make the study visit outside this interval.

<sup>&</sup>lt;sup>2</sup> Subjects may not be eligible for inclusion in the ATP cohort for analysis of immunogenicity and efficacy if they make the study visit outside this interval.

<sup>&</sup>lt;sup>2</sup> Subjects may not be eligible for inclusion in the ATP cohort for analysis of immunogenicity and efficacy if they make the study visit outside this interval.

205081 (MALARIA-092) Statistical Analysis Plan Final

The following group names will be used for the statistical analyses:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | AduFx | RTS,S/AS01 <sub>B</sub> full dose administered at Month 0, Month 1 and RTS,S/AS01 <sub>B</sub> 1/5 <sup>th</sup> dose administered at Month 7 |
| 2 | 2PedFx | RTS,S/AS01 <sub>E</sub> double dose administered at Month 0, Month 1 and double dose RTS,S/AS01 <sub>E</sub> 1/5 <sup>th</sup> dose administered at Month 7 |
| 3 | PedFx | RTS,S/AS01 <sub>E</sub> full dose administered at Month 0, Month 1 and RTS,S/AS01 <sub>E</sub> 1/5 <sup>th</sup> dose administered at Month 7 |
| 4 | Adu2Fx | RTS,S/AS01 <sub>B</sub> full dose at Month 0 and RTS,S/AS01 <sub>B</sub> 1/5 <sup>th</sup> dose administered at Month 1, Month 7 |
| 4 | Adu1Fx | RTS,S/AS01 <sub>B</sub> full dose at Month 0 and RTS,S/AS01 <sub>B</sub> 1/5 <sup>th</sup> dose administered at Month 7 |
| 5 | Control | Subjects will not receive any immunization but will undergo sporozoite challenge |

# Two defined pooled groups:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | Р | All subjects who have not been infected by <i>P. falciparum</i> parasitemia (defined by a positive blood slide) during the challenge and were part of one of the vaccinated groups |
| 2 | NP | All subjects who have been infected by <i>P. falciparum</i> parasitemia (defined by a positive blood slide) during the challenge and were part of one of the vaccinated groups |

## 3. OBJECTIVES

# 3.1. Primary objective

# 3.1.1. Efficacy

• To assess the vaccine efficacy against the occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) for each vaccination schedule (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx) versus the infectivity controls.

Refer to Section 4.1 for the definition of the primary endpoint.

# 3.2. Secondary objectives

# 3.2.1. Efficacy

- To assess the time to onset of *P. falciparum* parasitemia (defined by a positive blood slide) for each vaccination schedule (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx) versus the infectivity controls.
- To assess the occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) after vaccine administration for alternative vaccination schedules (2PedFx, PedFx, Adu2Fx, and Adu1Fx) versus the immunization schedule of reference (AduFx).
- To assess the time to onset of *P. falciparum* parasitemia (defined by a positive blood slide) after vaccine administration for alternative vaccination schedules (2PedFx, PedFx, Adu2Fx, and Adu1Fx) versus the immunization schedule of reference (AduFx).

## 3.2.2. Immunogenicity

For each vaccination schedule:

- To evaluate anti-CS repeat region antibody response at specified timepoints.
- To evaluate anti-HBs immunoglobulin G (IgG) antibody response at specified timepoints.

#### 3.2.3. Safety

For each vaccination schedule:

• To assess the safety (unsolicited AEs/AEs of specific interest/serious adverse events [SAEs]) and reactogenicity (solicited AEs).

Refer to Section 4.2 for the definition of the secondary endpoints.

# 3.3. Tertiary objectives

## 3.3.1. Immunogenicity

For each vaccination schedule:

- To evaluate anti-CS repeat region IgG avidity index at specified timepoints.
- To evaluate anti-full length CS protein IgG concentrations and anti-C terminal portion of the protein (C-term) IgG concentrations at specified timepoints.
- To evaluate anti-full length CS protein and anti-C-term IgG avidity at specified timepoints.

Note: other immuno-assays evaluating the immune response targeting the CS and HBsAg might be performed.

Refer to Section 4.3 for the definition of the tertiary endpoints.

#### 4. ENDPOINTS

# 4.1. Primary endpoint

# 4.1.1. Efficacy

- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>B</sub> administered as full doses at Month 0 and Month 1 and 1/5<sup>th</sup> dose at Month 7 (AduFx group) versus infectivity controls.
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>E</sub> administered as double dose at Month 0 and Month 1 and double 1/5<sup>th</sup> dose at Month 7 (2PedFx group) versus infectivity controls.
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>E</sub> administered as full doses at Month 0 and Month 1 and 1/5<sup>th</sup> dose at Month 7 (PedFx group) versus infectivity controls.
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>B</sub> administered as one full dose at Month 0 and 1/5<sup>th</sup> doses at Month 1 and Month 7 (Adu2Fx group) versus infectivity controls.
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>B</sub> administered as one full dose at Month 0 and 1/5<sup>th</sup> doses at Month 7 (Adu1Fx group) versus infectivity controls.

# 4.2. Secondary endpoints

# 4.2.1. Efficacy

- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>E</sub> administered as double dose at Month 0 and Month 1 and double 1/5<sup>th</sup> dose at Month 7 (2PedFx group) versus immunization schedule of reference (AduFx group).
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>E</sub> administered as full doses at Month 0 and Month 1 and 1/5<sup>th</sup> dose at Month 7 (PedFx) versus immunization schedule of reference (AduFx group).
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>B</sub> administered as one full dose at Month 0 and 1/5<sup>th</sup> full dose at Month 1 and Month 7 (Adu2Fx) versus immunization schedule of reference (AduFx group).
- Occurrence of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge, comparing RTS,S/AS01<sub>B</sub> administered as one full dose at Month 0 and 1/5<sup>th</sup> full doses at Month 7 (Adu1Fx) versus immunization schedule of reference (AduFx group).
- Time to onset of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge in each vaccination schedule versus immunization schedule of reference (AduFx group).
- Time to onset of *P. falciparum* parasitemia (defined by a positive blood slide) following sporozoite challenge in each vaccination schedule versus infectivity controls.

# 4.2.2. Immunogenicity

- For each vaccination schedule, the immune response to the CS antigen of the investigational vaccine:
  - Anti-CS repeat region antibody concentrations before vaccine administration (Day 0), one month post-Dose 2 (Day 58), six months post-Dose 2 (Day 196), one month post-Dose 3 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx groups and before vaccine administration (Day 0), before Dose 2 (Day 196), one month post-Dose 2 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from Adu1Fx group.

- For each vaccination schedule, the immune response to the hepatitis B antigen of the investigational vaccine:
  - Anti-HBs IgG antibody concentrations before vaccine administration (Day 0), one month post-Dose 2 (Day 58), six months post-Dose 2 (Day 196), one month post-Dose 3 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx groups and before vaccine administration (Day 0), before Dose 2 (Day 196), one month post-Dose 2 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from Adu1Fx group.

# 4.2.3. Safety

- Safety and reactogenicity of the investigational vaccine for each vaccination schedule:
  - Occurrence of solicited local and general AEs within seven days (day of vaccination and six subsequent days) after each vaccination.
  - Occurrence of unsolicited AEs within 30 days (day of vaccination and 29 subsequent days) after each vaccination, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification.
  - Occurrence of AEs within 30 days (day of challenge and 29 subsequent days) after challenge, according to the MedDRA classification.
  - Occurrence of SAEs (all, fatal, related to investigational vaccine) within 30 days (day of vaccination and 29 subsequent days) after each vaccination, according to the MedDRA classification.
  - Occurrence of SAEs (all, fatal, related to investigational vaccine) during the whole study period (from Dose 1 [Day 0] up to study conclusion [Day 376]), according to the MedDRA classification.
  - Occurrence of AEs and SAEs leading to withdrawal from further vaccination from Dose 1 (Day 0) up to study conclusion (Day 376), according to the MedDRA classification, for each vaccinated subject.
  - Occurrence of pIMDs from Dose 1 (Day 0) up to study conclusion (Day 376),
     according to the MedDRA classification, for each vaccinated subject.
  - Occurrence of meningitis from Dose 1 (Day 0) up to study conclusion (Day 376), according to the MedDRA classification, for each vaccinated subject.
  - Occurrence of abnormal laboratory values at screening, Day 35, Day 58, Day 203, Day 226, the day of first parasitemia, and Day 314 for each vaccinated subject and at screening, the day of first parasitemia and Day 314 for the infectivity control subjects.

- Safety after sporozoite challenge in the infectivity control group.
  - Occurrence of AEs within 30 days (day of challenge and 29 subsequent days) after challenge, according to the MedDRA classification.
  - Occurrence of SAEs (all, fatal, related) from day of challenge (Day 286) to the end of the challenge phase (Day 314), according to the MedDRA classification.

# 4.3. Tertiary endpoints

### 4.3.1. Immunogenicity

- For each vaccination schedule, the immune response to the CS antigen of the investigational vaccine:
  - Anti-CS repeat region IgG avidity index before vaccine administration (Day 0), one month post-Dose 2 (Day 58), six months post-Dose 2 (Day 196), one month post-Dose 3 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx groups and before vaccine administration (Day 0), before Dose 2 (Day 196), one month post-Dose 2 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from Adu1Fx group.
  - Anti-full length CS protein IgG concentrations and anti-C-term IgG concentrations before vaccine administration (Day 0), one month post-Dose 2 (Day 58), six months post-Dose 2 (Day 196), one month post-Dose 3 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx groups and before vaccine administration (Day 0), before Dose 2 (Day 196), one month post-Dose 2 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from Adu1Fx group.
  - Anti-full length CS protein and anti-C-term IgG avidity before vaccine administration (Day 0), one month post-Dose 2 (Day 58), six months post-Dose 2 (Day 196), one month post-Dose 3 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx groups and before vaccine administration (Day 0), before Dose 2 (Day 196), one month post-Dose 2 (Day 226), on the day of challenge (Day 286), 28 days post-challenge (Day 314), and at study end (Day 376) for subjects from Adu1Fx group.

Note: other immuno-assays evaluating the immune response targeting the CS and HBsAg might be performed.

## 5. ANALYSIS SETS

#### 5.1. Definition

Note that in order to align to ICH and CDISC terminology the According To Protocol (ATP) cohort has been renamed the Per-Protocol Set (PPS).

#### 5.1.1. Enrolled Set

The Enrolled Set will include all screened subjects who provide informed consent and provide demographic and/or other baseline screening measurements, regardless of the subject's randomization and vaccination status in the trial, and receive a subject ID.

# 5.1.2. Intent-to-treat set (ITTS)

The Intent-To-Treat Set (ITTS) will include all subjects who received at least one dose of study vaccine. The ITTS analysis will be performed per treatment actually administered. All challenged infectivity controls will also be included and will be presented as a separate study group.

# 5.1.3. Per-Protocol Set for analysis of immunogenicity and efficacy (PPS for analysis of immunogenicity and efficacy)

The PPS for analysis of immunogenicity and efficacy will include all subjects included in the ITTS who fulfilled all eligibility criteria and received all vaccinations according to protocol procedures within the protocol specified intervals, did not use any medication, vaccine or blood products forbidden by the protocol, did not report any underlying medical condition influencing the efficacy response, had available data concerning immunogenicity endpoint measures, and underwent *P. falciparum* challenge. This will include subjects for whom assay results are available for antibodies against at least one study vaccine antigen after vaccination.

# 5.1.4. Adapted Per-Protocol Set for analysis of efficacy (Adapted PPS for analysis of efficacy)

The Adapted PPS for analysis of efficacy will include all subjects included in the ITTS who fulfilled all eligibility criteria and received all vaccinations according to protocol procedures within the protocol specified intervals and underwent *P. falciparum* challenge.

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

#### 5.2.1. Elimination from ITTS

Code 1030 (Study vaccine not administered at all) for all subjects except those from the infectivity control group and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ITTS.

# 5.2.2. Elimination from the PPS for analysis of immunogenicity and efficacy

## 5.2.2.1. Excluded subjects

A subject will be excluded from the PPS analysis of immunogenicity and efficacy analysis under the following conditions

| Code | Condition under which the code is used |
|---|---|
| 900 | Invalid informed consent or fraud data |
| 1030 | Study vaccine not administered at all |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol |
| | Any investigational or non-registered vaccine other than the study vaccines used during the study period. |
| | A vaccine not foreseen by the study protocol administered during<br>the period starting seven days before each dose and ending seven<br>days after each dose of vaccines administration. |
| 1070 | Vaccination not according to protocol |
| | Incomplete vaccination course before treatment withdrawal or subject study conclusion. |
| | Administration not according to protocol for reason specified by the investigator, other than side, site and route. |
| | Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number). |
| | Study vaccine RTS,S/AS01 not prepared as per protocol |
| 1080 | Good Manufacturing Practice No-Go: Vaccine temperature deviation |
| 1090 | Expired vaccine administered |
| 2010 | Protocol violation (inclusion/exclusion criteria) |
| | Eligibility criteria not met with an impact on immunogenicity data |

205081 (MALARIA-092) Statistical Analysis Plan Final

| 1 | Otatistical Artalysis Flati Final |
|---|---|
| Code | Condition under which the code is used |
| 2040 | Administration of any medication forbidden by the protocol which may influence the efficacy endpoints |
| | Any investigational or non-registered product drug other than the study vaccines used during the study period. |
| | • Immunosuppressants or other immune-modifying drugs administered chronically (i.e. more than 14 days in total) during the study period. For corticosteroids, this will mean prednisone ≥ 20 mg/day (for adult subjects), or equivalent. Inhaled and topical steroids are allowed. |
| | Long-acting immune-modifying drugs administered at any time during the study period (e.g. infliximab). |
| | Immunoglobulins and/or any blood products administered during the study period. |
| | • Drugs known to have anti- <i>Plasmodium</i> properties, used during the challenge period before identification of parasitemia. |
| 2050 | Underlying medical condition forbidden by the protocol which may influence the efficacy endpoints |
| 2080 | Subjects did not comply with vaccination schedule |
| | (See Table 1, Table 2, Table 3) |
| 2090 | Subjects did not comply with blood sampling schedule |
| | (See Table 1, Table 2, Table 3) |
| 2100 | Serological results not available for anti-CS at all post-vaccination visits |
| 2120 | Obvious incoherence or abnormality or error in immunogenicity (antibody) data |
| 3000 | Subject did not undergo challenge |

# 5.2.3. Elimination from the Adapted PPS for analysis of efficacy

# 5.2.3.1. Excluded subjects

A subject will be excluded from the Adapted PPS analysis of efficacy analysis under the following conditions:

| Code | Condition under which the code is used |
|---|---|
| 900 | Invalid informed consent or fraud data |
| 1030 | Study vaccine not administered at all |
| 1070 | Vaccination not according to protocol |
| | Incomplete vaccination course before treatment withdrawal or subject study conclusion. |
| | Administration not according to protocol for reason specified by<br>the investigator, other than side, site and route. |
| | Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number). |
| | Study vaccine RTS,S/AS01 not prepared as per protocol |
| 3000 | Subject did not undergo challenge |

# 5.3. Important protocol deviations not leading to elimination from per-protocol analysis set

Important protocol deviations not leading to elimination from PPS are defined in MALARIA-092 (205081) Protocol Deviation Management Plan.

PPD

(MALARIA-092 (205081) Protocol Deviation Management Plan)

# 6. STATISTICAL ANALYSES

Note that standard data derivation rules and statistical methods are described in Annex 1 and will not be repeated below.

# 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

A study flow table (consort) will be generated to present the number of subjects screened, randomized, receiving doses and included in the PPS for analyses.

The analysis of demographics will be performed on the ITTS and on the PPS for analysis of immunogenicity and efficacy.

Demographic characteristics (age at first vaccination in years for the vaccinated groups and at the time of the screening for the control group, gender, and race) will be summarized by group and overall using descriptive statistics:

- Frequency tables will be generated for categorical variables such as race.
- Mean, median, standard deviation (SD) and range will be provided for continuous data such as age.

Withdrawal status will be summarized by group using descriptive statistics:

- The number of subjects enrolled into the study as well as the number of subjects excluded from PPS for analyses will be tabulated.
- The number of withdrawn subjects will be tabulated according to the reason for withdrawal.

# 6.2. Exposure

#### 6.2.1. Analysis of exposure planned in the protocol

The number and percentages of subjects with vaccination will be summarized overall and by group for all groups where a vaccination is part of the study procedure. The analysis of exposure will be performed on the ITTS.

# 6.3. Efficacy analysis

# 6.3.1. Analysis of efficacy planned in the protocol

The analysis of efficacy will be performed on the PPS for analysis of immunogenicity and efficacy.

Efficacy will be assessed by comparison of *P. falciparum* parasitemia incidence and time to onset of *P. falciparum* parasitemia after sporozoite challenge.

Vaccine efficacy (VE) is defined as 100\*(1-Relative Risk). Relative risk of infection and 95% CI will be calculated.

Fisher's Exact test will be used for the comparison of *P. falciparum* parasitemia incidence after challenge between each one of the vaccine groups (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx) and the infectivity control group.

Kaplan-Meier analysis will be performed on time to onset of *P. falciparum* parasitemia, for comparisons between each one of the vaccine groups (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx) and the infectivity control group, using the log-rank statistic.

The same methodology will be applied for the evaluation of the vaccinated groups versus the immunization schedule of reference (AduFx group).

All statistical tests will be two-tailed at 5% significance level.

#### 6.3.2. Additional considerations

#### 6.3.2.1. Case definition

The primary case definition of P. falciparum infection is an asexual blood stage P. falciparum parasite density > 0 detected by blood slide reading.

## 6.3.2.2. Risk periods

For the analyses of time to onset of parasitemia (Kaplan-Meier and Log-Rank), time at risk will start on first day of challenge. Time at risk will be censored on protocol visit D314 (28 days post challenge), drop-out date, start date of antimalarial treatment or date meeting an endpoint, whichever occurs first. Time at risk will be calculated as: censor date – date challenge + 1.

For the analysis of proportion affected (relative risk), all subjects included in the PPS for analysis of immunogenicity and efficacy will be considered at risk of infection and no censoring or elimination will be applied for subjects not completing the entire protocol defined post challenge follow-up (visit D314 - 28 days post challenge).

# 6.4. Immunogenicity analysis

# 6.4.1. Analysis of immunogenicity planned in the protocol

The analysis of immunogenicity will be performed on the PPS for analysis of immunogenicity and efficacy.

For each study group, at each timepoint that a blood sample result is available:

The percentage of subjects with seropositive levels of anti-CS (proportion of subjects with anti-CS antibody concentrations  $\geq 1.9$  EU/ml) with 95% CI will be determined at specified blood sampling timepoints in each group (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx). Anti-CS antibody concentrations will be summarized by GMC. Anti-CS antibody concentrations will be displayed using reverse cumulative curves. Similar analysis will be performed for the anti-full length CS protein (proportion of subjects with anti-CS antibody titres  $\geq 200$  1/DIL) and anti-C-term antibodies (proportion of subjects with anti-CS antibody concentrations  $\geq 100$  EPT).

The percentage of subjects with seroprotection levels of anti-HBs (anti-HBs antibody concentrations  $\geq 10$  mIU/ml) with 95% CI will be determined at specified blood sampling timepoints in each groups (AduFx, 2PedFx, PedFx, Adu2Fx, and Adu1Fx). Anti-HBs antibody concentrations will be summarized by GMC. Anti-HBs antibody concentrations will be displayed using reverse cumulative curves.

Anti-CS, anti-full length CS protein and anti-CS avidity index will be summarized by mean, SD, median and quartile and box and whiskers plots will be generated.

#### 6.4.2. Additional considerations

In addition to the previous analyses, the immunogenicity analyses will be performed per protection status (P and NP) overall (pooled vaccine groups) and within each vaccine group.

Exploratory analyses using logistic regression models will be evaluated to describe the relationship between immune read outs and the probability of infection (P vs NP). Explanatory variables will include all or a part of available immune read outs at time of analysis (anti-CS, anti-full length CS protein, avidity index).

In a first step, immune responses will be plotted by group and protection status as well as cross-tabulated to understand potential correlation structures. Then, relevant models will be constructed to evaluate what are the independent predictors of protection, both pooled over the treatment groups (is/are there a generic driver(s)?) and by treatment schedule/including interactions (is protection mediated through different mechanisms between schedules?).

# 6.5. Analysis of safety

# 6.5.1. Analysis of safety planned in the protocol

The analysis of safety will be performed on the ITTS.

The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the 7-day or 30 day follow-up period after each vaccine dose and overall will be tabulated with exact 95% CI. The percentage of doses followed by at least one local AE (solicited and unsolicited), by at least one general AE (solicited and unsolicited) and by any AE during the 7-day or 30-day follow-up period will be tabulated with exact 95% CI. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination and for any Grade 3 AEs considered related to vaccination.

The percentage of subjects reporting each individual solicited local AE (any grade and Grade 3) and each individual solicited general AE (any grade, Grade 3, any related, Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period (Day 0-6) after each vaccine dose and overall will be tabulated for each group. Similarly, the percentage of doses followed by each individual solicited local and general AE will be tabulated, for the overall and for each vaccination course, with exact 95% CI.

For fever (fever is defined as temperature  $\geq 37.5^{\circ}\text{C}/99.5^{\circ}\text{F}$  for oral, axillary or tympanic route, or  $\geq 38.0^{\circ}\text{C}/100.4^{\circ}\text{F}$  for rectal route), the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the first seven days (Day 0-6) after each vaccine dose and overall will be tabulated. Similar tabulations will be performed for any fever with a causal relationship to vaccination and Grade 3 (> 39.0°C) causally related fever. The maximum temperature reported over the 7-day follow-up period (Day 0-6) overall doses will be tabulated.

The percentage of subjects reporting unsolicited AEs within 30 days (Day 0-29) after each vaccine dose (overall doses) and percentage of subjects reporting AEs after the sporozoite challenge will be tabulated by group and by MedDRA preferred term with exact 95% CI. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs and for Grade 3 causally related unsolicited AEs.

The percentage of subjects reporting SAEs (all, fatal, related) occurring within 30 days (day of vaccination and 29 subsequent days) after each dose of study vaccine, classified by the MedDRA preferred term level will be tabulated with exact 95% CI.

The percentage of subjects reporting SAEs (all, fatal, related) occurring from Dose 1 (Day 0) until last study visit (Day 376), classified by the MedDRA preferred term level will be tabulated with exact 95% CI.

The percentage of subjects reporting SAEs (all, fatal, related) occurring from day of challenge (Day 286) to the end of the challenge phase (Day 314), according to the MedDRA classification will be tabulated with exact 95% CI.

205081 (MALARIA-092) Statistical Analysis Plan Final

Subjects reporting pregnancies will be described.

The percentage of subjects reporting an AE or SAE leading to withdrawal from further vaccination from Dose 1 (Day 0) until last study visit (Day 376), classified by MedDRA preferred term level, will be tabulated with exact 95% CI.

The percentage of vaccinated subjects reporting AEs of specific interest (meningitis and pIMDs) from Dose 1 (Day 0) until last study visit (Day 376), classified by MedDRA preferred term level, will be tabulated with exact 95% CI.

Biochemistry (ALT, AST and creatinine) and hematological (hemoglobin, WBC and platelets) laboratory values will be presented by visit according to toxicity grading scales and tabulated by group.

The normal ranges and toxicity grading for laboratory safety parameters used in this study are presented in Table 4

## Table 4 Toxicity grading scales for blood testing

| Adverse event | Intensity grade | Intensity* |
|---|---|---|
| Hemoglobin (males) | Normal range | ≥12.5 g/dl |
| | 1 | < 12.5 but ≥ 11.0 g/dl |
| | 2 | < 11.0 but ≥ 10.0 g/dl |
| | 3 | < 10.0 g/dl |
| Hemoglobin (females) | Normal range | ≥11.5 g/dl |
| | 1 | < 11.5 but ≥ 10.5 g/dl |
| | 2 | < 10.5 but ≥ 9.5 g/dl |
| | 3 | < 9.5 g/dl |
| Increase in leukocytes | Normal range | ≤10799 cells/mm <sup>3</sup> |
| (WBC) | 1 | 10800 - 15000 cells/mm <sup>3</sup> |
| , | 2 | 15001 - 20000 cells/mm <sup>3</sup> |
| | 3 | > 20001 cells/mm <sup>3</sup> |
| Decrease in leukocytes | Normal range | ≥3200 cells/mm <sup>3</sup> |
| (WBC) | 1 | 2500 - 3199 cells/mm <sup>3</sup> |
| , | 2 | 1500 - 2499 cells/mm <sup>3</sup> |
| | 3 | < 1500 cells/mm <sup>3</sup> |
| Decrease in platelets | Normal | ≥140000 cells/mm <sup>3</sup> |
| · | 1 | 125000 - 139000 cells/mm <sup>3</sup> |
| | 2 | 100000 - 124000 cells/mm <sup>3</sup> |
| | 3 | < 100000 cells/mm <sup>3</sup> |
| Alanine Aminotransferase | Normal range | Below ULN (60 U/I for males; 40 U/I for females) |
| | 1 | 1.1 - 2.5 x ULN |
| | 2 | 2.6 – 5 x ULN |
| | 3 | > 5 x ULN |
| Aspartate Aminotransferase | Normal range | Below ULN (40 U/I for males; 35 U/I for females) |
| | 1 | 1.1 - 2.5 x ULN |
| | 2 | 2.6 – 5 x ULN |
| | 3 | > 5 x ULN |
| Creatinine (males) | Normal range | ≤1.39 mg/dl |
| | 1 | 1.4 - 1.79 mg/dl |
| | 2 | 1.8 - 2.0 mg/dl |
| | 3 | > 2.0 mg/dl |
| Creatinine (females) | Normal range | ≤1.29 mg/dl |
| | 1 | 1.3 – 1.69 mg/dl |
| | 2 | 1.7 – 1.9 mg/dl |
| I II Alexandra Back of a consol as | 3 | >1.9 mg/dl |

ULN: upper limit of normal range

The percentage of subjects using concomitant medication (any medication, any antipyretic and any prophylactic medication, respectively) during the 7-day follow-up period (Day 0-6) after vaccination will be summarized by group after each dose and overall. The percentage of subjects using concomitant medication during the entire sporozoite challenge (D286-314) will be summarized by group.

<sup>\*</sup> Grading scale adapted from [FDA guidance for industry toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (September 2007)].

#### 6.5.2. Additional considerations

A summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes:

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| FATIGUE | 10016256 | Fatigue |
| FEVER | 10016558 | Fever |
| GASTROINTESTINAL | 10017944 | Gastrointestinal disorder |
| HEADACHE | 10019211 | Headache |
| PAIN | 10022086 | Injection site pain |
| REDNESS | 10022098 | Redness at injection site |
| SWELLING | 10053425 | Swelling at injection site |

The following analysis will be performed if at least 5 subjects have used concomitant vaccination during the 7-day follow-up period (Day 0-6) after study vaccination during the full study period.

The percentage of subjects using any concomitant vaccination during the 7-day follow-up period (Day 0-6) after study vaccination will be summarized by group after each dose and overall. The percentage of subjects using concomitant vaccination during the entire sporozoite challenge will be summarized by group.

Note that the study will be converted in CDISC. Accordingly protocol Day 0-Day N will be replaced by Day 1-Day N+1 for the statistical analysis.

## 7. ANALYSIS INTERPRETATION

All the analyses performed during this study will be descriptive.

### 8. CONDUCT OF ANALYSES

# 8.1. Sequence of analyses

The analyses will be performed stepwise:

- An interim analysis to allow an internal decision for the choice of the booster dose in study Malaria-102 will be performed as soon as the results of the challenge phase will be available on data as clean as possible. This analysis will be descriptive and performed on the Adapted PPS for analysis of efficacy.
- When all the remaining data up to Day 376 will be available, the main analysis will be performed. An integrated study report will be written.

# 8.2. Statistical considerations for interim analyses

A descriptive analysis to evaluate VE against infection of *P. falciparum* will be performed on the Adapted PPS for analysis of efficacy at the time of the interim analysis. Note that the main objective of the study linked to this endpoint will be analysed at the end of the study, on the PPS for analysis of immunogenicity and efficacy and can output different results.

# 9. CHANGES FROM PLANNED ANALYSES

The Total vaccinated cohort (TVC) defined in the protocol has been replaced by the Intent-To-Treat Set (ITTS) to include both subjects vaccinated and subjects from the infectivity control group in the same cohort.

An interim analysis has been added to allow an internal decision for the choice of the booster dose in study Malaria-102. This analysis will be descriptive and performed on data as cleaned as possible.

To allow an interim analysis as close as possible to the main analysis, an Adapted PPS for analysis of efficacy has been created.

An analysis of concomitant vaccination has been added to assess any effect on immune response or safety.

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS, Annex). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulations of individual data such as listings of SAEs. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day & month are missing, 30 June is used.
- Onset day for an event (AE, medication, vaccination): The onset day is the number of days between the last study vaccination & the onset/start date of the event. This is 1 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.
- Duration: Duration of an event is expressed in days. It is the number of days between the start & the stop dates + 1. Therefore duration is 1 day for an event starting & ending on the same day.

#### 11.2.2. Dose number

- The study dose number is defined in reference to the number of study visits at which vaccination occurred. More specifically dose 1 refers to all vaccines administered at the first vaccination visit while dose 2 corresponds to all vaccinations administered at the second vaccination visit even if this is the first time a product is administered to the subject.
- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an AE begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose. In case a study dose is not administered (eg dose 2) and an event occurs after the subsequent study dose (eg 3rd study dose), the relative dose of the event will be study dose associated to the subsequent study dose (eg dose 3).
- The number of doses for a product is the number of times the product was administered to a subject.
- The incidence per dose is the number of vaccination visits at which an event was reported among all vaccination visits.

### 11.2.3. Demography

- Age: Age at the reference activity, computed as the number of years between the date of birth and the reference activity. Note that due to incomplete date, the derived age may be incorrect by 1 year when month is missing from the birthdate. This may lead to an apparent inconsistency between the derived age and the eligibility criteria/the age category used for randomization.
- Conversion of weight to kg

The following conversion rule is used:

Weight in Kilogrammes= weight in Pounds / 2.2 + weight in Ounces / 35.2

The result is rounded to 2 decimals.

• Conversion of height to cm

The following conversion rule is used:

Height in Centimetres = Height in Feet \* 30.48 + Height in Inches \* 2.54

The result is rounded to the unit (ie no decimal).

• Conversion of temperature to °C

The following conversion rule is used:

- Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

# 11.2.4. Immunogenicity

- For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.
- The Geometric Mean Concentrations (GMCs) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMC calculation. The cut-off value is defined by the laboratory before the analysis.
- The percentage of subjects seropositive/seroprotected and associated two-sided 95% Clopper-Pearson confidence intervals (CIs) will be computed by vaccine group for each available immunogenicity monitoring.
- A subject seropositive for anti-CS antibody will be a subject whose antibody concentration will be greater than or equal to the cut-off value (anti-CS ≥ 1.9 EU/ml).
- Seroprotection rate for anti-HBs antibody is defined as the percentage of subjects with antibody concentration greater than or equal to an established cut-off (anti-HBs ≥ 10 mIU/ml).

### 11.2.5. Safety

- Handling of missing data: subjects who missed reporting symptoms (unsolicited or concomitant medications) will be treated as subjects without symptoms (unsolicited or concomitant medications, respectively). In case of significant non-compliance of study procedures for reporting symptoms, the analysis plan will be reassessed to ensure more accurate reporting of study data by further analysis.
- For the analysis of solicited symptoms, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the ES will include only subjects/doses with documented safety data (i.e. symptom screen/sheet completed).
- For a given subject and the analysis of solicited symptoms within 7 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the ES will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed). More specifically the following rules will be used:
  - Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
  - Subjects who documented the presence of a solicited symptom and fully or
    partially recorded daily measurement over the solicited period will be included
    in the summaries at that dose and classified according to their maximum
    observed daily recording over the solicited period.
  - Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be assigned to the lowest intensity category at that dose (i.e., 37.5°C for fever or grade 1 for other symptoms).
  - Doses without symptom sheets documented will be excluded.
- For analysis of unsolicited AEs, such as SAEs or AEs by primary MedDRA term, and for the analysis of concomitant medications, all vaccinated subjects will be considered.
- For the analysis, temperatures will be coded as follows:

| Grade | Temperature |
|-------|--------------------------------------------|
| 0 | < 37.5°C (< 99.5°F) |
| 1 | ≥ 37.5°C (≥ 99.5°F) to ≤ 38.0°C (100.4°F) |
| 2 | > 38.0°C (> 100.4°F) to ≤ 39.0°C (102.1°F) |
| 3 | > 39.0°C (102.1°F) |

• For the analysis, local injection site redness and swelling will be coded as follows:

| Grade | Temperature |
|-------|---------------------|
| 0 | 0 mm |
| 1 | > 0 to ≤ 50 mm |
| 2 | > 50 mm to ≤ 100 mm |
| 3 | > 100 mm |

205081 (MALARIA-092) Statistical Analysis Plan Final

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for<br>Vaccination phase | N used for deriving % per dose for<br>Vaccination phase |
|---|---|---|
| Concomitant vaccination | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Solicited general symptom | All subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) | All study visits with study vaccine administered and with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) |
| Solicited local symptom | All subjects with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) | All study visits with study vaccine administered and with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) |
| Unsolicited symptom | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered | All study visits with study vaccine administered |

• Related dose: The related dose for an event (e.g., AE, medication, vaccination,...) is the study dose given before an event. In case the event takes place on a day a study dose is given, if the investigator has indicated the timing (before or after the vaccination) the related dose for this event is the most recent study dose given before this event. If the investigator has not indicated the timing, the related dose will be that of the study dose even if the event actually took place before.

#### Number of decimals displayed:

The following decimal description from the decision rules will be used for demography, efficacy, immunogenicity and safety/reactogenicity results.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| Demographic characteristics | Mean, median age | 1 |
| Demographic characteristics | SD (age) | 1 |
| Reactogenicity | Mean, Min, Q1, Median, Q3, Max for duration | 1 |
| All summaries | % of count, including LL & UL of CI | 1 |
| All summaries | p-value | 3 |